CLINICAL TRIAL: NCT00539487
Title: TOP -Study Telmisartan - Therapy of Hypertension and Life-style Changes in Cardiovascular Risk Patients
Brief Title: Observational Non-interventional Study (Anwendungsbeobachtung) With Telmisartan in High-risk Hypertensives
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 502.523
Record Dates: First submitted 2007-09-25; First posted 2007-10-04 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Hypertension; Obesity
MeSH Terms: conditions — Hypertension; Obesity

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This observational non-interventional study will assess (under conditions of clinical practice in daily routine) the antihypertensive efficacy of telmisartan treatment with or without active promotion of lifestyle changes in hypertensive patients at high cardiovascular risk

DETAILED DESCRIPTION:
Study Design:

ELIGIBILITY:
Inclusion Criteria:

patients with essential hypertension aged >/= 18 years with one of the following risk factors: history of coronary artery disease or stroke/TIA or peripheral artery disease or diabetes mellitus.

Exclusion Criteria:

according to SPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hypertensive patients
Sampling Method: Non-Probability Sample
Enrollment: 5827 (Actual)
Dates: Start 2007-01; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Blood pressure reduction | 4 month

SECONDARY OUTCOMES:
Change in metabolic parameters Safety

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2389):
- Germany (2389):
  - Boehringer Ingelheim Investigational Site 1, Aachen
  - Boehringer Ingelheim Investigational Site 2, Aachen
  - Boehringer Ingelheim Investigational Site 3, Aachen
  - Boehringer Ingelheim Investigational Site 4, Aachen
  - Boehringer Ingelheim Investigational Site 5, Aachen
  - Boehringer Ingelheim Investigational Site 6, Aachen
  - Boehringer Ingelheim Investigational Site 7, Aachen
  - Boehringer Ingelheim Investigational Site 8, Aachen
  - Boehringer Ingelheim Investigational Site, Aalen
  - Boehringer Ingelheim Investigational Site, Aarbergen
  - Boehringer Ingelheim Investigational Site, Abstatt
  - Boehringer Ingelheim Investigational Site, Achern
  - Boehringer Ingelheim Investigational Site 1, Adendorf
  - Boehringer Ingelheim Investigational Site 2, Adendorf
  - Boehringer Ingelheim Investigational Site 3, Adendorf
  - Boehringer Ingelheim Investigational Site, Aham
  - Boehringer Ingelheim Investigational Site 1, Ahaus
  - Boehringer Ingelheim Investigational Site 2, Ahaus
  - Boehringer Ingelheim Investigational Site, Ahlen
  - Boehringer Ingelheim Investigational Site, Ahorn
  - Boehringer Ingelheim Investigational Site, Ahorntal
  - Boehringer Ingelheim Investigational Site, Ahrensbök
  - Boehringer Ingelheim Investigational Site, Ahrensburg
  - Boehringer Ingelheim Investigational Site, Ahrensfelde
  - Boehringer Ingelheim Investigational Site, Aichach
  - Boehringer Ingelheim Investigational Site, Aichtal
  - Boehringer Ingelheim Investigational Site, Ainring
  - Boehringer Ingelheim Investigational Site, Albbruck
  - Boehringer Ingelheim Investigational Site 1, Albstadt
  - Boehringer Ingelheim Investigational Site 2, Albstadt
  - Boehringer Ingelheim Investigational Site 3, Albstadt
  - Boehringer Ingelheim Investigational Site 4, Albstadt
  - Boehringer Ingelheim Investigational Site, Aldenhoven
  - Boehringer Ingelheim Investigational Site, Alfeld
  - Boehringer Ingelheim Investigational Site, Algermissen
  - Boehringer Ingelheim Investigational Site, Allendorf
  - Boehringer Ingelheim Investigational Site, Allmendingen
  - Boehringer Ingelheim Investigational Site 1, Alpen
  - Boehringer Ingelheim Investigational Site 2, Alpen
  - Boehringer Ingelheim Investigational Site, Alsdorf
  - Boehringer Ingelheim Investigational Site, Altena
  - Boehringer Ingelheim Investigational Site 1, Altenburg
  - Boehringer Ingelheim Investigational Site 2, Altenburg
  - Boehringer Ingelheim Investigational Site 1, Altenholz
  - Boehringer Ingelheim Investigational Site 2, Altenholz
  - Boehringer Ingelheim Investigational Site 3, Altenholz
  - Boehringer Ingelheim Investigational Site 1, Altenstadt
  - Boehringer Ingelheim Investigational Site 2, Altenstadt
  - Boehringer Ingelheim Investigational Site, Altensteig
  - Boehringer Ingelheim Investigational Site, Altlußheim
  - Boehringer Ingelheim Investigational Site, Altmittweida
  - Boehringer Ingelheim Investigational Site, Altötting
  - Boehringer Ingelheim Investigational Site, Altrip
  - Boehringer Ingelheim Investigational Site, Alzenau in Unterfranken
  - Boehringer Ingelheim Investigational Site, Amberg
  - Boehringer Ingelheim Investigational Site, Ammerbuch
  - Boehringer Ingelheim Investigational Site, Anklam
  - Boehringer Ingelheim Investigational Site, Ansbach
  - Boehringer Ingelheim Investigational Site, Apelern
  - Boehringer Ingelheim Investigational Site 1, Apolda
  - Boehringer Ingelheim Investigational Site 2, Apolda
  - Boehringer Ingelheim Investigational Site, Appenweier
  - Boehringer Ingelheim Investigational Site, Arenshausen
  - Boehringer Ingelheim Investigational Site, Artern
  - Boehringer Ingelheim Investigational Site 1, Arzberg
  - Boehringer Ingelheim Investigational Site 2, Arzberg
  - Boehringer Ingelheim Investigational Site, Aschaffenburg
  - Boehringer Ingelheim Investigational Site 1, Aschersleben
  - Boehringer Ingelheim Investigational Site 2, Aschersleben
  - Boehringer Ingelheim Investigational Site, Aspach
  - Boehringer Ingelheim Investigational Site, Attendorn
  - Boehringer Ingelheim Investigational Site, Attenkirchen
  - Boehringer Ingelheim Investigational Site, Auerbach
  - Boehringer Ingelheim Investigational Site 1, Augsburg
  - Boehringer Ingelheim Investigational Site 2, Augsburg
  - Boehringer Ingelheim Investigational Site 3, Augsburg
  - Boehringer Ingelheim Investigational Site 4, Augsburg
  - Boehringer Ingelheim Investigational Site 5, Augsburg
  - Boehringer Ingelheim Investigational Site, Auw
  - Boehringer Ingelheim Investigational Site 1, Aßlar
  - Boehringer Ingelheim Investigational Site 2, Aßlar
  - Boehringer Ingelheim Investigational Site, Baar-Ebenhausen
  - Boehringer Ingelheim Investigational Site, Babenhausen
  - Boehringer Ingelheim Investigational Site 1, Backnang
  - Boehringer Ingelheim Investigational Site 2, Backnang
  - Boehringer Ingelheim Investigational Site 3, Backnang
  - Boehringer Ingelheim Investigational Site 1, Bad Bentheim
  - Boehringer Ingelheim Investigational Site 2, Bad Bentheim
  - Boehringer Ingelheim Investigational Site, Bad Berka
  - Boehringer Ingelheim Investigational Site, Bad Bevensen
  - Boehringer Ingelheim Investigational Site, Bad Blankenburg
  - Boehringer Ingelheim Investigational Site, Bad Doberan
  - Boehringer Ingelheim Investigational Site 1, Bad Düben
  - Boehringer Ingelheim Investigational Site 2, Bad Düben
  - Boehringer Ingelheim Investigational Site, Bad Dürrenberg
  - Boehringer Ingelheim Investigational Site, Bad Dürrheim
  - Boehringer Ingelheim Investigational Site 1, Bad Elster
  - Boehringer Ingelheim Investigational Site 2, Bad Elster
  - Boehringer Ingelheim Investigational Site, Bad Ems
  - Boehringer Ingelheim Investigational Site, Bad Essen
  - Boehringer Ingelheim Investigational Site, Bad Fallingbostel
  - Boehringer Ingelheim Investigational Site 1, Bad Frankenhausen
  - Boehringer Ingelheim Investigational Site 2, Bad Frankenhausen
  - Boehringer Ingelheim Investigational Site, Bad Freienwalde
  - Boehringer Ingelheim Investigational Site 1, Bad Kissingen
  - Boehringer Ingelheim Investigational Site 2, Bad Kissingen
  - Boehringer Ingelheim Investigational Site, Bad Krozingen
  - Boehringer Ingelheim Investigational Site, Bad Laasphe
  - Boehringer Ingelheim Investigational Site, Bad Laer
  - Boehringer Ingelheim Investigational Site, Bad Langensalza
  - Boehringer Ingelheim Investigational Site, Bad Lausick
  - Boehringer Ingelheim Investigational Site 1, Bad Lauterberg im Harz
  - Boehringer Ingelheim Investigational Site 2, Bad Lauterberg im Harz
  - Boehringer Ingelheim Investigational Site, Bad Marienberg
  - Boehringer Ingelheim Investigational Site, Bad Mergentheim
  - Boehringer Ingelheim Investigational Site, Bad Münstereifel
  - Boehringer Ingelheim Investigational Site 1, Bad Nenndorf
  - Boehringer Ingelheim Investigational Site 2, Bad Nenndorf
  - Boehringer Ingelheim Investigational Site, Bad Neustadt an der Saale
  - Boehringer Ingelheim Investigational Site 1, Bad Oeynhausen
  - Boehringer Ingelheim Investigational Site 2, Bad Oeynhausen
  - Boehringer Ingelheim Investigational Site, Bad Rappenau
  - Boehringer Ingelheim Investigational Site, Bad Reichenhall
  - Boehringer Ingelheim Investigational Site, Bad Sachsa
  - Boehringer Ingelheim Investigational Site 1, Bad Salzuflen
  - Boehringer Ingelheim Investigational Site 2, Bad Salzuflen
  - Boehringer Ingelheim Investigational Site 3, Bad Salzuflen
  - Boehringer Ingelheim Investigational Site 4, Bad Salzuflen
  - Boehringer Ingelheim Investigational Site 1, Bad Salzungen
  - Boehringer Ingelheim Investigational Site 2, Bad Salzungen
  - Boehringer Ingelheim Investigational Site 3, Bad Salzungen
  - Boehringer Ingelheim Investigational Site, Bad Schandau
  - Boehringer Ingelheim Investigational Site, Bad Schönborn
  - Boehringer Ingelheim Investigational Site 1, Bad Schussenried
  - Boehringer Ingelheim Investigational Site 2, Bad Schussenried
  - Boehringer Ingelheim Investigational Site 3, Bad Schussenried
  - Boehringer Ingelheim Investigational Site 1, Bad Schwartau
  - Boehringer Ingelheim Investigational Site 2, Bad Schwartau
  - Boehringer Ingelheim Investigational Site, Bad Sulza
  - Boehringer Ingelheim Investigational Site, Bad Tennstedt
  - Boehringer Ingelheim Investigational Site, Bad Tölz
  - Boehringer Ingelheim Investigational Site, Bad Vilbel
  - Boehringer Ingelheim Investigational Site, Bad Waldsee
  - Boehringer Ingelheim Investigational Site, Bad Wilsnack
  - Boehringer Ingelheim Investigational Site, Bad Wörishofen
  - Boehringer Ingelheim Investigational Site, Badel
  - Boehringer Ingelheim Investigational Site 1, Baden-Baden
  - Boehringer Ingelheim Investigational Site 2, Baden-Baden
  - Boehringer Ingelheim Investigational Site, Bahrdorf
  - Boehringer Ingelheim Investigational Site, Baienfurt
  - Boehringer Ingelheim Investigational Site, Bakum
  - Boehringer Ingelheim Investigational Site, Ballenstedt
  - Boehringer Ingelheim Investigational Site 1, Bamberg
  - Boehringer Ingelheim Investigational Site 2, Bamberg
  - Boehringer Ingelheim Investigational Site 3, Bamberg
  - Boehringer Ingelheim Investigational Site, Bandelin
  - Boehringer Ingelheim Investigational Site 1, Barchfeld
  - Boehringer Ingelheim Investigational Site 2, Barchfeld
  - Boehringer Ingelheim Investigational Site, Barmstedt
  - Boehringer Ingelheim Investigational Site, Barsbüttel
  - Boehringer Ingelheim Investigational Site, Barsinghausen
  - Boehringer Ingelheim Investigational Site, Barth
  - Boehringer Ingelheim Investigational Site, Barßel
  - Boehringer Ingelheim Investigational Site, Baunatal
  - Boehringer Ingelheim Investigational Site 1, Bautzen
  - Boehringer Ingelheim Investigational Site 2, Bautzen
  - Boehringer Ingelheim Investigational Site 3, Bautzen
  - Boehringer Ingelheim Investigational Site, Bayreuth
  - Boehringer Ingelheim Investigational Site, Bärnau
  - Boehringer Ingelheim Investigational Site, Bechtheim
  - Boehringer Ingelheim Investigational Site, Beckum
  - Boehringer Ingelheim Investigational Site, Beeskow
  - Boehringer Ingelheim Investigational Site, Belm
  - Boehringer Ingelheim Investigational Site, Bensheim
  - Boehringer Ingelheim Investigational Site, Berching
  - Boehringer Ingelheim Investigational Site, Berchtesgaden
  - Boehringer Ingelheim Investigational Site 1, Bergfelde
  - Boehringer Ingelheim Investigational Site 2, Bergfelde
  - Boehringer Ingelheim Investigational Site 1, Bergheim
  - Boehringer Ingelheim Investigational Site 2, Bergheim
  - Boehringer Ingelheim Investigational Site 1, Bergisch Gladbach
  - Boehringer Ingelheim Investigational Site 2, Bergisch Gladbach
  - Boehringer Ingelheim Investigational Site 3, Bergisch Gladbach
  - Boehringer Ingelheim Investigational Site 4, Bergisch Gladbach
  - Boehringer Ingelheim Investigational Site 1, Bergkamen
  - Boehringer Ingelheim Investigational Site 2, Bergkamen
  - Boehringer Ingelheim Investigational Site 1, Bergrheinfeld
  - Boehringer Ingelheim Investigational Site 2, Bergrheinfeld
  - Boehringer Ingelheim Investigational Site 10, Berlin
  - Boehringer Ingelheim Investigational Site 11, Berlin
  - Boehringer Ingelheim Investigational Site 12, Berlin
  - Boehringer Ingelheim Investigational Site 13, Berlin
  - Boehringer Ingelheim Investigational Site 14, Berlin
  - Boehringer Ingelheim Investigational Site 15, Berlin
  - Boehringer Ingelheim Investigational Site 16, Berlin
  - Boehringer Ingelheim Investigational Site 17, Berlin
  - Boehringer Ingelheim Investigational Site 18, Berlin
  - Boehringer Ingelheim Investigational Site 19, Berlin
  - Boehringer Ingelheim Investigational Site 1, Berlin
  - Boehringer Ingelheim Investigational Site 20, Berlin
  - Boehringer Ingelheim Investigational Site 21, Berlin
  - Boehringer Ingelheim Investigational Site 22, Berlin
  - Boehringer Ingelheim Investigational Site 23, Berlin
  - Boehringer Ingelheim Investigational Site 24, Berlin
  - Boehringer Ingelheim Investigational Site 25, Berlin
  - Boehringer Ingelheim Investigational Site 26, Berlin
  - Boehringer Ingelheim Investigational Site 27, Berlin
  - Boehringer Ingelheim Investigational Site 28, Berlin
  - Boehringer Ingelheim Investigational Site 29, Berlin
  - Boehringer Ingelheim Investigational Site 2, Berlin
  - Boehringer Ingelheim Investigational Site 30, Berlin
  - Boehringer Ingelheim Investigational Site 31, Berlin
  - Boehringer Ingelheim Investigational Site 32, Berlin
  - Boehringer Ingelheim Investigational Site 33, Berlin
  - Boehringer Ingelheim Investigational Site 34, Berlin
  - Boehringer Ingelheim Investigational Site 35, Berlin
  - Boehringer Ingelheim Investigational Site 36, Berlin
  - Boehringer Ingelheim Investigational Site 37, Berlin
  - Boehringer Ingelheim Investigational Site 38, Berlin
  - Boehringer Ingelheim Investigational Site 39, Berlin
  - Boehringer Ingelheim Investigational Site 3, Berlin
  - Boehringer Ingelheim Investigational Site 40, Berlin
  - Boehringer Ingelheim Investigational Site 41, Berlin
  - Boehringer Ingelheim Investigational Site 42, Berlin
  - Boehringer Ingelheim Investigational Site 43, Berlin
  - Boehringer Ingelheim Investigational Site 44, Berlin
  - Boehringer Ingelheim Investigational Site 45, Berlin
  - Boehringer Ingelheim Investigational Site 46, Berlin
  - Boehringer Ingelheim Investigational Site 47, Berlin
  - Boehringer Ingelheim Investigational Site 48, Berlin
  - Boehringer Ingelheim Investigational Site 49, Berlin
  - Boehringer Ingelheim Investigational Site 4, Berlin
  - Boehringer Ingelheim Investigational Site 50, Berlin
  - Boehringer Ingelheim Investigational Site 51, Berlin
  - Boehringer Ingelheim Investigational Site 52, Berlin
  - Boehringer Ingelheim Investigational Site 53, Berlin
  - Boehringer Ingelheim Investigational Site 54, Berlin
  - Boehringer Ingelheim Investigational Site 55, Berlin
  - Boehringer Ingelheim Investigational Site 56, Berlin
  - Boehringer Ingelheim Investigational Site 57, Berlin
  - Boehringer Ingelheim Investigational Site 58, Berlin
  - Boehringer Ingelheim Investigational Site 59, Berlin
  - Boehringer Ingelheim Investigational Site 5, Berlin
  - Boehringer Ingelheim Investigational Site 60, Berlin
  - Boehringer Ingelheim Investigational Site 61, Berlin
  - Boehringer Ingelheim Investigational Site 62, Berlin
  - Boehringer Ingelheim Investigational Site 63, Berlin
  - Boehringer Ingelheim Investigational Site 64, Berlin
  - Boehringer Ingelheim Investigational Site 65, Berlin
  - Boehringer Ingelheim Investigational Site 66, Berlin
  - Boehringer Ingelheim Investigational Site 67, Berlin
  - Boehringer Ingelheim Investigational Site 68, Berlin
  - Boehringer Ingelheim Investigational Site 69, Berlin
  - Boehringer Ingelheim Investigational Site 6, Berlin
  - Boehringer Ingelheim Investigational Site 70, Berlin
  - Boehringer Ingelheim Investigational Site 71, Berlin
  - Boehringer Ingelheim Investigational Site 72, Berlin
  - Boehringer Ingelheim Investigational Site 73, Berlin
  - Boehringer Ingelheim Investigational Site 74, Berlin
  - Boehringer Ingelheim Investigational Site 75, Berlin
  - Boehringer Ingelheim Investigational Site 76, Berlin
  - Boehringer Ingelheim Investigational Site 77, Berlin
  - Boehringer Ingelheim Investigational Site 78, Berlin
  - Boehringer Ingelheim Investigational Site 79, Berlin
  - Boehringer Ingelheim Investigational Site 7, Berlin
  - Boehringer Ingelheim Investigational Site 80, Berlin
  - Boehringer Ingelheim Investigational Site 81, Berlin
  - Boehringer Ingelheim Investigational Site 82, Berlin
  - Boehringer Ingelheim Investigational Site 83, Berlin
  - Boehringer Ingelheim Investigational Site 84, Berlin
  - Boehringer Ingelheim Investigational Site 85, Berlin
  - Boehringer Ingelheim Investigational Site 86, Berlin
  - Boehringer Ingelheim Investigational Site 87, Berlin
  - Boehringer Ingelheim Investigational Site 88, Berlin
  - Boehringer Ingelheim Investigational Site 89, Berlin
  - Boehringer Ingelheim Investigational Site 8, Berlin
  - Boehringer Ingelheim Investigational Site 90, Berlin
  - Boehringer Ingelheim Investigational Site 91, Berlin
  - Boehringer Ingelheim Investigational Site 92, Berlin
  - Boehringer Ingelheim Investigational Site 93, Berlin
  - Boehringer Ingelheim Investigational Site 9, Berlin
  - Boehringer Ingelheim Investigational Site 1, Bernau
  - Boehringer Ingelheim Investigational Site 2, Bernau
  - Boehringer Ingelheim Investigational Site, Bernau
  - Boehringer Ingelheim Investigational Site 1, Bernburg
  - Boehringer Ingelheim Investigational Site 2, Bernburg
  - Boehringer Ingelheim Investigational Site 3, Bernburg
  - Boehringer Ingelheim Investigational Site, Bernhardswald
  - Boehringer Ingelheim Investigational Site 1, Bernsdorf
  - Boehringer Ingelheim Investigational Site 2, Bernsdorf
  - Boehringer Ingelheim Investigational Site, Besigheim
  - Boehringer Ingelheim Investigational Site, Bestwig
  - Boehringer Ingelheim Investigational Site, Beucha
  - Boehringer Ingelheim Investigational Site, Bevern
  - Boehringer Ingelheim Investigational Site 1, Biberach
  - Boehringer Ingelheim Investigational Site 2, Biberach
  - Boehringer Ingelheim Investigational Site 3, Biberach
  - Boehringer Ingelheim Investigational Site, Biblis
  - Boehringer Ingelheim Investigational Site, Biedenkopf
  - Boehringer Ingelheim Investigational Site 1, Bielefeld
  - Boehringer Ingelheim Investigational Site 2, Bielefeld
  - Boehringer Ingelheim Investigational Site 3, Bielefeld
  - Boehringer Ingelheim Investigational Site, Bienenbüttel
  - Boehringer Ingelheim Investigational Site 1, Bietigheim-Bissingen
  - Boehringer Ingelheim Investigational Site 2, Bietigheim-Bissingen
  - Boehringer Ingelheim Investigational Site 3, Bietigheim-Bissingen
  - Boehringer Ingelheim Investigational Site 4, Bietigheim-Bissingen
  - Boehringer Ingelheim Investigational Site, Bindlach
  - Boehringer Ingelheim Investigational Site 1, Bingen
  - Boehringer Ingelheim Investigational Site 2, Bingen
  - Boehringer Ingelheim Investigational Site, Birkenau
  - Boehringer Ingelheim Investigational Site, Bischofferode
  - Boehringer Ingelheim Investigational Site 1, Bischofsheim
  - Boehringer Ingelheim Investigational Site 2, Bischofsheim
  - Boehringer Ingelheim Investigational Site, Blankenhain
  - Boehringer Ingelheim Investigational Site, Blaustein
  - Boehringer Ingelheim Investigational Site, Bleckede
  - Boehringer Ingelheim Investigational Site, Bobenheim-Roxheim
  - Boehringer Ingelheim Investigational Site, Bobritzsch
  - Boehringer Ingelheim Investigational Site 1, Bocholt
  - Boehringer Ingelheim Investigational Site 2, Bocholt
  - Boehringer Ingelheim Investigational Site 3, Bocholt
  - Boehringer Ingelheim Investigational Site 10, Bochum
  - Boehringer Ingelheim Investigational Site 11, Bochum
  - Boehringer Ingelheim Investigational Site 12, Bochum
  - Boehringer Ingelheim Investigational Site 13, Bochum
  - Boehringer Ingelheim Investigational Site 1, Bochum
  - Boehringer Ingelheim Investigational Site 2, Bochum
  - Boehringer Ingelheim Investigational Site 3, Bochum
  - Boehringer Ingelheim Investigational Site 4, Bochum
  - Boehringer Ingelheim Investigational Site 5, Bochum
  - Boehringer Ingelheim Investigational Site 6, Bochum
  - Boehringer Ingelheim Investigational Site 7, Bochum
  - Boehringer Ingelheim Investigational Site 8, Bochum
  - Boehringer Ingelheim Investigational Site 9, Bochum
  - Boehringer Ingelheim Investigational Site, Bockenem
  - Boehringer Ingelheim Investigational Site 1, Bodenwerder
  - Boehringer Ingelheim Investigational Site 2, Bodenwerder
  - Boehringer Ingelheim Investigational Site, Bogen
  - Boehringer Ingelheim Investigational Site 1, Bonn
  - Boehringer Ingelheim Investigational Site 2, Bonn
  - Boehringer Ingelheim Investigational Site 3, Bonn
  - Boehringer Ingelheim Investigational Site 4, Bonn
  - Boehringer Ingelheim Investigational Site, Boostedt
  - Boehringer Ingelheim Investigational Site 1, Bopfingen
  - Boehringer Ingelheim Investigational Site 2, Bopfingen
  - Boehringer Ingelheim Investigational Site, Boppard
  - Boehringer Ingelheim Investigational Site 1, Bornheim
  - Boehringer Ingelheim Investigational Site 2, Bornheim
  - Boehringer Ingelheim Investigational Site 1, Bottrop
  - Boehringer Ingelheim Investigational Site 2, Bottrop
  - Boehringer Ingelheim Investigational Site 3, Bottrop
  - Boehringer Ingelheim Investigational Site, Bovenden
  - Boehringer Ingelheim Investigational Site 1, Böblingen
  - Boehringer Ingelheim Investigational Site 2, Böblingen
  - Boehringer Ingelheim Investigational Site, Böhlen
  - Boehringer Ingelheim Investigational Site, Bönen
  - Boehringer Ingelheim Investigational Site, Brackenheim
  - Boehringer Ingelheim Investigational Site, Brake
  - Boehringer Ingelheim Investigational Site, Brakel
  - Boehringer Ingelheim Investigational Site 1, Brandenburg
  - Boehringer Ingelheim Investigational Site 2, Brandenburg
  - Boehringer Ingelheim Investigational Site 3, Brandenburg
  - Boehringer Ingelheim Investigational Site 4, Brandenburg
  - Boehringer Ingelheim Investigational Site 1, Braunschweig
  - Boehringer Ingelheim Investigational Site 2, Braunschweig
  - Boehringer Ingelheim Investigational Site 3, Braunschweig
  - Boehringer Ingelheim Investigational Site 4, Braunschweig
  - Boehringer Ingelheim Investigational Site 5, Braunschweig
  - Boehringer Ingelheim Investigational Site 6, Braunschweig
  - Boehringer Ingelheim Investigational Site, Brechen
  - Boehringer Ingelheim Investigational Site, Bredstedt
  - Boehringer Ingelheim Investigational Site, Brehna
  - Boehringer Ingelheim Investigational Site, Breitenbach
  - Boehringer Ingelheim Investigational Site 1, Bremen
  - Boehringer Ingelheim Investigational Site 2, Bremen
  - Boehringer Ingelheim Investigational Site 3, Bremen
  - Boehringer Ingelheim Investigational Site 4, Bremen
  - Boehringer Ingelheim Investigational Site 5, Bremen
  - Boehringer Ingelheim Investigational Site 6, Bremen
  - Boehringer Ingelheim Investigational Site 7, Bremen
  - Boehringer Ingelheim Investigational Site 8, Bremen
  - Boehringer Ingelheim Investigational Site 1, Bremerhaven
  - Boehringer Ingelheim Investigational Site 2, Bremerhaven
  - Boehringer Ingelheim Investigational Site 3, Bremerhaven
  - Boehringer Ingelheim Investigational Site, Brensbach
  - Boehringer Ingelheim Investigational Site, Bretten
  - Boehringer Ingelheim Investigational Site 1, Breuberg
  - Boehringer Ingelheim Investigational Site 2, Breuberg
  - Boehringer Ingelheim Investigational Site, Brieselang
  - Boehringer Ingelheim Investigational Site, Broderstorf
  - Boehringer Ingelheim Investigational Site, Bruchsal
  - Boehringer Ingelheim Investigational Site, Bruckmühl
  - Boehringer Ingelheim Investigational Site, Brücken
  - Boehringer Ingelheim Investigational Site, Brüggen
  - Boehringer Ingelheim Investigational Site 1, Brühl
  - Boehringer Ingelheim Investigational Site 2, Brühl
  - Boehringer Ingelheim Investigational Site 3, Brühl
  - Boehringer Ingelheim Investigational Site 1, Buchbach
  - Boehringer Ingelheim Investigational Site 2, Buchbach
  - Boehringer Ingelheim Investigational Site, Buchholz
  - Boehringer Ingelheim Investigational Site, Burg
  - Boehringer Ingelheim Investigational Site 1, Burghausen
  - Boehringer Ingelheim Investigational Site 2, Burghausen
  - Boehringer Ingelheim Investigational Site, Burgstall
  - Boehringer Ingelheim Investigational Site, Burgstädt
  - Boehringer Ingelheim Investigational Site, Burgstetten
  - Boehringer Ingelheim Investigational Site, Burow
  - Boehringer Ingelheim Investigational Site, Butzbach
  - Boehringer Ingelheim Investigational Site, Büchen
  - Boehringer Ingelheim Investigational Site, Bülkau
  - Boehringer Ingelheim Investigational Site 1, Bünde
  - Boehringer Ingelheim Investigational Site 2, Bünde
  - Boehringer Ingelheim Investigational Site 3, Bünde
  - Boehringer Ingelheim Investigational Site, Büren
  - Boehringer Ingelheim Investigational Site, Calbe
  - Boehringer Ingelheim Investigational Site, Camburg
  - Boehringer Ingelheim Investigational Site, Carlsberg
  - Boehringer Ingelheim Investigational Site 1, Castrop-Rauxel
  - Boehringer Ingelheim Investigational Site 2, Castrop-Rauxel
  - Boehringer Ingelheim Investigational Site 3, Castrop-Rauxel
  - Boehringer Ingelheim Investigational Site 4, Castrop-Rauxel
  - Boehringer Ingelheim Investigational Site 5, Castrop-Rauxel
  - Boehringer Ingelheim Investigational Site 6, Castrop-Rauxel
  - Boehringer Ingelheim Investigational Site 1, Celle
  - Boehringer Ingelheim Investigational Site 2, Celle
  - Boehringer Ingelheim Investigational Site 3, Celle
  - Boehringer Ingelheim Investigational Site 4, Celle
  - Boehringer Ingelheim Investigational Site 10, Chemnitz
  - Boehringer Ingelheim Investigational Site 11, Chemnitz
  - Boehringer Ingelheim Investigational Site 12, Chemnitz
  - Boehringer Ingelheim Investigational Site 13, Chemnitz
  - Boehringer Ingelheim Investigational Site 14, Chemnitz
  - Boehringer Ingelheim Investigational Site 15, Chemnitz
  - Boehringer Ingelheim Investigational Site 16, Chemnitz
  - Boehringer Ingelheim Investigational Site 17, Chemnitz
  - Boehringer Ingelheim Investigational Site 18, Chemnitz
  - Boehringer Ingelheim Investigational Site 1, Chemnitz
  - Boehringer Ingelheim Investigational Site 2, Chemnitz
  - Boehringer Ingelheim Investigational Site 3, Chemnitz
  - Boehringer Ingelheim Investigational Site 4, Chemnitz
  - Boehringer Ingelheim Investigational Site 5, Chemnitz
  - Boehringer Ingelheim Investigational Site 6, Chemnitz
  - Boehringer Ingelheim Investigational Site 7, Chemnitz
  - Boehringer Ingelheim Investigational Site 8, Chemnitz
  - Boehringer Ingelheim Investigational Site 9, Chemnitz
  - Boehringer Ingelheim Investigational Site, Claußnitz
  - Boehringer Ingelheim Investigational Site, Cloppenburg
  - Boehringer Ingelheim Investigational Site, Coburg
  - Boehringer Ingelheim Investigational Site, Colditz
  - Boehringer Ingelheim Investigational Site 10, Cologne
  - Boehringer Ingelheim Investigational Site 11, Cologne
  - Boehringer Ingelheim Investigational Site 12, Cologne
  - Boehringer Ingelheim Investigational Site 13, Cologne
  - Boehringer Ingelheim Investigational Site 14, Cologne
  - Boehringer Ingelheim Investigational Site 15, Cologne
  - Boehringer Ingelheim Investigational Site 16, Cologne
  - Boehringer Ingelheim Investigational Site 17, Cologne
  - Boehringer Ingelheim Investigational Site 18, Cologne
  - Boehringer Ingelheim Investigational Site 19, Cologne
  - Boehringer Ingelheim Investigational Site 1, Cologne
  - Boehringer Ingelheim Investigational Site 20, Cologne
  - Boehringer Ingelheim Investigational Site 21, Cologne
  - Boehringer Ingelheim Investigational Site 22, Cologne
  - Boehringer Ingelheim Investigational Site 23, Cologne
  - Boehringer Ingelheim Investigational Site 24, Cologne
  - Boehringer Ingelheim Investigational Site 25, Cologne
  - Boehringer Ingelheim Investigational Site 26, Cologne
  - Boehringer Ingelheim Investigational Site 27, Cologne
  - Boehringer Ingelheim Investigational Site 2, Cologne
  - Boehringer Ingelheim Investigational Site 3, Cologne
  - Boehringer Ingelheim Investigational Site 4, Cologne
  - Boehringer Ingelheim Investigational Site 5, Cologne
  - Boehringer Ingelheim Investigational Site 6, Cologne
  - Boehringer Ingelheim Investigational Site 7, Cologne
  - Boehringer Ingelheim Investigational Site 8, Cologne
  - Boehringer Ingelheim Investigational Site 9, Cologne
  - Boehringer Ingelheim Investigational Site, Coppenbrügge
  - Boehringer Ingelheim Investigational Site 1, Cottbus
  - Boehringer Ingelheim Investigational Site 2, Cottbus
  - Boehringer Ingelheim Investigational Site 3, Cottbus
  - Boehringer Ingelheim Investigational Site 1, Crivitz
  - Boehringer Ingelheim Investigational Site 2, Crivitz
  - Boehringer Ingelheim Investigational Site, Dabel
  - Boehringer Ingelheim Investigational Site, Dachau
  - Boehringer Ingelheim Investigational Site 1, Darmstadt
  - Boehringer Ingelheim Investigational Site 2, Darmstadt
  - Boehringer Ingelheim Investigational Site 3, Darmstadt
  - Boehringer Ingelheim Investigational Site 1, Datteln
  - Boehringer Ingelheim Investigational Site 2, Datteln
  - Boehringer Ingelheim Investigational Site, Daun
  - Boehringer Ingelheim Investigational Site, Dautphetal
  - Boehringer Ingelheim Investigational Site, Deggendorf
  - Boehringer Ingelheim Investigational Site, Deidesheim
  - Boehringer Ingelheim Investigational Site 1, Delitzsch
  - Boehringer Ingelheim Investigational Site 2, Delitzsch
  - Boehringer Ingelheim Investigational Site, Delligsen
  - Boehringer Ingelheim Investigational Site 1, Delmenhorst
  - Boehringer Ingelheim Investigational Site 2, Delmenhorst
  - Boehringer Ingelheim Investigational Site 3, Delmenhorst
  - Boehringer Ingelheim Investigational Site, Derenburg
  - Boehringer Ingelheim Investigational Site, Dernbach
  - Boehringer Ingelheim Investigational Site, Dersekow
  - Boehringer Ingelheim Investigational Site, Dersum
  - Boehringer Ingelheim Investigational Site 1, Dessau
  - Boehringer Ingelheim Investigational Site 2, Dessau
  - Boehringer Ingelheim Investigational Site 3, Dessau
  - Boehringer Ingelheim Investigational Site 1, Detmold
  - Boehringer Ingelheim Investigational Site 2, Detmold
  - Boehringer Ingelheim Investigational Site 3, Detmold
  - Boehringer Ingelheim Investigational Site 4, Detmold
  - Boehringer Ingelheim Investigational Site 5, Detmold
  - Boehringer Ingelheim Investigational Site, Dettingen
  - Boehringer Ingelheim Investigational Site, Diepholz
  - Boehringer Ingelheim Investigational Site 1, Dierdorf
  - Boehringer Ingelheim Investigational Site 2, Dierdorf
  - Boehringer Ingelheim Investigational Site, Dietzenbach
  - Boehringer Ingelheim Investigational Site, Diez
  - Boehringer Ingelheim Investigational Site, Dillenburg
  - Boehringer Ingelheim Investigational Site 1, Dillingen
  - Boehringer Ingelheim Investigational Site 2, Dillingen
  - Boehringer Ingelheim Investigational Site 3, Dillingen
  - Boehringer Ingelheim Investigational Site 4, Dillingen
  - Boehringer Ingelheim Investigational Site, Dingolfing
  - Boehringer Ingelheim Investigational Site, Dinkelsbühl
  - Boehringer Ingelheim Investigational Site 1, Dinslaken
  - Boehringer Ingelheim Investigational Site 2, Dinslaken
  - Boehringer Ingelheim Investigational Site 3, Dinslaken
  - Boehringer Ingelheim Investigational Site, Doberschütz
  - Boehringer Ingelheim Investigational Site, Dollern
  - Boehringer Ingelheim Investigational Site, Dormagen
  - Boehringer Ingelheim Investigational Site, Dorn-Dürkheim
  - Boehringer Ingelheim Investigational Site, Dornburg
  - Boehringer Ingelheim Investigational Site 1, Dorsten
  - Boehringer Ingelheim Investigational Site 2, Dorsten
  - Boehringer Ingelheim Investigational Site 3, Dorsten
  - Boehringer Ingelheim Investigational Site 10, Dortmund
  - Boehringer Ingelheim Investigational Site 11, Dortmund
  - Boehringer Ingelheim Investigational Site 12, Dortmund
  - Boehringer Ingelheim Investigational Site 13, Dortmund
  - Boehringer Ingelheim Investigational Site 14, Dortmund
  - Boehringer Ingelheim Investigational Site 15, Dortmund
  - Boehringer Ingelheim Investigational Site 16, Dortmund
  - Boehringer Ingelheim Investigational Site 17, Dortmund
  - Boehringer Ingelheim Investigational Site 18, Dortmund
  - Boehringer Ingelheim Investigational Site 19, Dortmund
  - Boehringer Ingelheim Investigational Site 1, Dortmund
  - Boehringer Ingelheim Investigational Site 20, Dortmund
  - Boehringer Ingelheim Investigational Site 21, Dortmund
  - Boehringer Ingelheim Investigational Site 22, Dortmund
  - Boehringer Ingelheim Investigational Site 23, Dortmund
  - Boehringer Ingelheim Investigational Site 24, Dortmund
  - Boehringer Ingelheim Investigational Site 25, Dortmund
  - Boehringer Ingelheim Investigational Site 2, Dortmund
  - Boehringer Ingelheim Investigational Site 3, Dortmund
  - Boehringer Ingelheim Investigational Site 4, Dortmund
  - Boehringer Ingelheim Investigational Site 5, Dortmund
  - Boehringer Ingelheim Investigational Site 6, Dortmund
  - Boehringer Ingelheim Investigational Site 7, Dortmund
  - Boehringer Ingelheim Investigational Site 8, Dortmund
  - Boehringer Ingelheim Investigational Site 9, Dortmund
  - Boehringer Ingelheim Investigational Site, Dossenheim
  - Boehringer Ingelheim Investigational Site, Döbeln
  - Boehringer Ingelheim Investigational Site, Dörentrup
  - Boehringer Ingelheim Investigational Site, Dörzbach
  - Boehringer Ingelheim Investigational Site, Dreetz
  - Boehringer Ingelheim Investigational Site 1, Dreieich
  - Boehringer Ingelheim Investigational Site 2, Dreieich
  - Boehringer Ingelheim Investigational Site, Drensteinfurt
  - Boehringer Ingelheim Investigational Site 10, Dresden
  - Boehringer Ingelheim Investigational Site 11, Dresden
  - Boehringer Ingelheim Investigational Site 12, Dresden
  - Boehringer Ingelheim Investigational Site 13, Dresden
  - Boehringer Ingelheim Investigational Site 14, Dresden
  - Boehringer Ingelheim Investigational Site 15, Dresden
  - Boehringer Ingelheim Investigational Site 16, Dresden
  - Boehringer Ingelheim Investigational Site 17, Dresden
  - Boehringer Ingelheim Investigational Site 18, Dresden
  - Boehringer Ingelheim Investigational Site 19, Dresden
  - Boehringer Ingelheim Investigational Site 1, Dresden
  - Boehringer Ingelheim Investigational Site 20, Dresden
  - Boehringer Ingelheim Investigational Site 21, Dresden
  - Boehringer Ingelheim Investigational Site 22, Dresden
  - Boehringer Ingelheim Investigational Site 23, Dresden
  - Boehringer Ingelheim Investigational Site 2, Dresden
  - Boehringer Ingelheim Investigational Site 3, Dresden
  - Boehringer Ingelheim Investigational Site 4, Dresden
  - Boehringer Ingelheim Investigational Site 5, Dresden
  - Boehringer Ingelheim Investigational Site 6, Dresden
  - Boehringer Ingelheim Investigational Site 7, Dresden
  - Boehringer Ingelheim Investigational Site 8, Dresden
  - Boehringer Ingelheim Investigational Site 9, Dresden
  - Boehringer Ingelheim Investigational Site 10, Duisburg
  - Boehringer Ingelheim Investigational Site 11, Duisburg
  - Boehringer Ingelheim Investigational Site 12, Duisburg
  - Boehringer Ingelheim Investigational Site 13, Duisburg
  - Boehringer Ingelheim Investigational Site 14, Duisburg
  - Boehringer Ingelheim Investigational Site 15, Duisburg
  - Boehringer Ingelheim Investigational Site 16, Duisburg
  - Boehringer Ingelheim Investigational Site 1, Duisburg
  - Boehringer Ingelheim Investigational Site 2, Duisburg
  - Boehringer Ingelheim Investigational Site 3, Duisburg
  - Boehringer Ingelheim Investigational Site 4, Duisburg
  - Boehringer Ingelheim Investigational Site 5, Duisburg
  - Boehringer Ingelheim Investigational Site 6, Duisburg
  - Boehringer Ingelheim Investigational Site 7, Duisburg
  - Boehringer Ingelheim Investigational Site 8, Duisburg
  - Boehringer Ingelheim Investigational Site 9, Duisburg
  - Boehringer Ingelheim Investigational Site 1, Durmersheim
  - Boehringer Ingelheim Investigational Site 2, Durmersheim
  - Boehringer Ingelheim Investigational Site 10, Düsseldorf
  - Boehringer Ingelheim Investigational Site 11, Düsseldorf
  - Boehringer Ingelheim Investigational Site 12, Düsseldorf
  - Boehringer Ingelheim Investigational Site 13, Düsseldorf
  - Boehringer Ingelheim Investigational Site 14, Düsseldorf
  - Boehringer Ingelheim Investigational Site 15, Düsseldorf
  - Boehringer Ingelheim Investigational Site 16, Düsseldorf
  - Boehringer Ingelheim Investigational Site 17, Düsseldorf
  - Boehringer Ingelheim Investigational Site 18, Düsseldorf
  - Boehringer Ingelheim Investigational Site 19, Düsseldorf
  - Boehringer Ingelheim Investigational Site 1, Düsseldorf
  - Boehringer Ingelheim Investigational Site 20, Düsseldorf
  - Boehringer Ingelheim Investigational Site 21, Düsseldorf
  - Boehringer Ingelheim Investigational Site 22, Düsseldorf
  - Boehringer Ingelheim Investigational Site 23, Düsseldorf
  - Boehringer Ingelheim Investigational Site 2, Düsseldorf
  - Boehringer Ingelheim Investigational Site 3, Düsseldorf
  - Boehringer Ingelheim Investigational Site 4, Düsseldorf
  - Boehringer Ingelheim Investigational Site 5, Düsseldorf
  - Boehringer Ingelheim Investigational Site 6, Düsseldorf
  - Boehringer Ingelheim Investigational Site 7, Düsseldorf
  - Boehringer Ingelheim Investigational Site 8, Düsseldorf
  - Boehringer Ingelheim Investigational Site 9, Düsseldorf
  - Boehringer Ingelheim Investigational Site, Ebeleben
  - Boehringer Ingelheim Investigational Site, Eberbach
  - Boehringer Ingelheim Investigational Site, Ebergötzen
  - Boehringer Ingelheim Investigational Site, Ebersbach
  - Boehringer Ingelheim Investigational Site, Ebersdorf
  - Boehringer Ingelheim Investigational Site, Eberstadt
  - Boehringer Ingelheim Investigational Site 1, Eberswalde
  - Boehringer Ingelheim Investigational Site 2, Eberswalde
  - Boehringer Ingelheim Investigational Site, Eckernförde
  - Boehringer Ingelheim Investigational Site, Edertal
  - Boehringer Ingelheim Investigational Site, Edling
  - Boehringer Ingelheim Investigational Site 1, Eggenstein-Leopoldshafen
  - Boehringer Ingelheim Investigational Site 2, Eggenstein-Leopoldshafen
  - Boehringer Ingelheim Investigational Site 1, Ehingen
  - Boehringer Ingelheim Investigational Site 2, Ehingen
  - Boehringer Ingelheim Investigational Site, Ehra-Lessien
  - Boehringer Ingelheim Investigational Site, Ehringshausen
  - Boehringer Ingelheim Investigational Site, Eibelstadt
  - Boehringer Ingelheim Investigational Site, Eilenburg
  - Boehringer Ingelheim Investigational Site, Eilsdorf
  - Boehringer Ingelheim Investigational Site, Eilsleben
  - Boehringer Ingelheim Investigational Site, Eisenach
  - Boehringer Ingelheim Investigational Site, Eisenberg
  - Boehringer Ingelheim Investigational Site 1, Eisenhüttenstadt
  - Boehringer Ingelheim Investigational Site 2, Eisenhüttenstadt
  - Boehringer Ingelheim Investigational Site, Eisleben Lutherstadt
  - Boehringer Ingelheim Investigational Site, Eislingen
  - Boehringer Ingelheim Investigational Site 1, Eitorf
  - Boehringer Ingelheim Investigational Site 2, Eitorf
  - Boehringer Ingelheim Investigational Site, Ellerstadt
  - Boehringer Ingelheim Investigational Site, Ellhofen
  - Boehringer Ingelheim Investigational Site 1, Elmshorn
  - Boehringer Ingelheim Investigational Site 2, Elmshorn
  - Boehringer Ingelheim Investigational Site, Elsterwerda
  - Boehringer Ingelheim Investigational Site, Elz
  - Boehringer Ingelheim Investigational Site, Elze
  - Boehringer Ingelheim Investigational Site, Emmendingen
  - Boehringer Ingelheim Investigational Site, Emmerich
  - Boehringer Ingelheim Investigational Site, Emmering
  - Boehringer Ingelheim Investigational Site, Emmerting
  - Boehringer Ingelheim Investigational Site, Emskirchen
  - Boehringer Ingelheim Investigational Site 1, Engelskirchen
  - Boehringer Ingelheim Investigational Site 2, Engelskirchen
  - Boehringer Ingelheim Investigational Site, Enger
  - Boehringer Ingelheim Investigational Site, Enkenbach-Alsenborn
  - Boehringer Ingelheim Investigational Site, Ennepetal
  - Boehringer Ingelheim Investigational Site, Ense
  - Boehringer Ingelheim Investigational Site, Eppelborn
  - Boehringer Ingelheim Investigational Site 1, Eppelheim
  - Boehringer Ingelheim Investigational Site 2, Eppelheim
  - Boehringer Ingelheim Investigational Site, Eppstein
  - Boehringer Ingelheim Investigational Site 1, Erbach im Odenwald
  - Boehringer Ingelheim Investigational Site 2, Erbach im Odenwald
  - Boehringer Ingelheim Investigational Site, Erding
  - Boehringer Ingelheim Investigational Site 1, Erftstadt
  - Boehringer Ingelheim Investigational Site 2, Erftstadt
  - Boehringer Ingelheim Investigational Site 10, Erfurt
  - Boehringer Ingelheim Investigational Site 11, Erfurt
  - Boehringer Ingelheim Investigational Site 1, Erfurt
  - Boehringer Ingelheim Investigational Site 2, Erfurt
  - Boehringer Ingelheim Investigational Site 3, Erfurt
  - Boehringer Ingelheim Investigational Site 4, Erfurt
  - Boehringer Ingelheim Investigational Site 5, Erfurt
  - Boehringer Ingelheim Investigational Site 6, Erfurt
  - Boehringer Ingelheim Investigational Site 7, Erfurt
  - Boehringer Ingelheim Investigational Site 8, Erfurt
  - Boehringer Ingelheim Investigational Site 9, Erfurt
  - Boehringer Ingelheim Investigational Site, Erkner
  - Boehringer Ingelheim Investigational Site, Erlangen
  - Boehringer Ingelheim Investigational Site, Erndtebrück
  - Boehringer Ingelheim Investigational Site, Eschershausen
  - Boehringer Ingelheim Investigational Site 1, Eschwege
  - Boehringer Ingelheim Investigational Site 2, Eschwege
  - Boehringer Ingelheim Investigational Site 1, Eschweiler
  - Boehringer Ingelheim Investigational Site 2, Eschweiler
  - Boehringer Ingelheim Investigational Site 3, Eschweiler
  - Boehringer Ingelheim Investigational Site 4, Eschweiler
  - Boehringer Ingelheim Investigational Site 5, Eschweiler
  - Boehringer Ingelheim Investigational Site 10, Essen
  - Boehringer Ingelheim Investigational Site 11, Essen
  - Boehringer Ingelheim Investigational Site 12, Essen
  - Boehringer Ingelheim Investigational Site 13, Essen
  - Boehringer Ingelheim Investigational Site 14, Essen
  - Boehringer Ingelheim Investigational Site 15, Essen
  - Boehringer Ingelheim Investigational Site 16, Essen
  - Boehringer Ingelheim Investigational Site 17, Essen
  - Boehringer Ingelheim Investigational Site 18, Essen
  - Boehringer Ingelheim Investigational Site 19, Essen
  - Boehringer Ingelheim Investigational Site 1, Essen
  - Boehringer Ingelheim Investigational Site 20, Essen
  - Boehringer Ingelheim Investigational Site 21, Essen
  - Boehringer Ingelheim Investigational Site 22, Essen
  - Boehringer Ingelheim Investigational Site 23, Essen
  - Boehringer Ingelheim Investigational Site 24, Essen
  - Boehringer Ingelheim Investigational Site 25, Essen
  - Boehringer Ingelheim Investigational Site 26, Essen
  - Boehringer Ingelheim Investigational Site 27, Essen
  - Boehringer Ingelheim Investigational Site 2, Essen
  - Boehringer Ingelheim Investigational Site 3, Essen
  - Boehringer Ingelheim Investigational Site 4, Essen
  - Boehringer Ingelheim Investigational Site 5, Essen
  - Boehringer Ingelheim Investigational Site 6, Essen
  - Boehringer Ingelheim Investigational Site 7, Essen
  - Boehringer Ingelheim Investigational Site 8, Essen
  - Boehringer Ingelheim Investigational Site 9, Essen
  - Boehringer Ingelheim Investigational Site 1, Esslingen am Neckar
  - Boehringer Ingelheim Investigational Site 2, Esslingen am Neckar
  - Boehringer Ingelheim Investigational Site 3, Esslingen am Neckar
  - Boehringer Ingelheim Investigational Site, Ettlingen
  - Boehringer Ingelheim Investigational Site, Euba
  - Boehringer Ingelheim Investigational Site, Eurasburg
  - Boehringer Ingelheim Investigational Site 1, Euskirchen
  - Boehringer Ingelheim Investigational Site 2, Euskirchen
  - Boehringer Ingelheim Investigational Site, Eutin
  - Boehringer Ingelheim Investigational Site, Extertal
  - Boehringer Ingelheim Investigational Site, Falkenberg
  - Boehringer Ingelheim Investigational Site, Falkensee
  - Boehringer Ingelheim Investigational Site, Faßberg
  - Boehringer Ingelheim Investigational Site, Fehrbellin
  - Boehringer Ingelheim Investigational Site, Fellbach
  - Boehringer Ingelheim Investigational Site 1, Felsberg
  - Boehringer Ingelheim Investigational Site 2, Felsberg
  - Boehringer Ingelheim Investigational Site, Fichtenberg
  - Boehringer Ingelheim Investigational Site, Filderstadt
  - Boehringer Ingelheim Investigational Site, Finnentrop
  - Boehringer Ingelheim Investigational Site, Finsterwalde
  - Boehringer Ingelheim Investigational Site, Flöha
  - Boehringer Ingelheim Investigational Site, Flörsheim
  - Boehringer Ingelheim Investigational Site, Flörsheim-Dalsheim
  - Boehringer Ingelheim Investigational Site, Forchheim
  - Boehringer Ingelheim Investigational Site 1, Forst
  - Boehringer Ingelheim Investigational Site 2, Forst
  - Boehringer Ingelheim Investigational Site 1, Frankenberg
  - Boehringer Ingelheim Investigational Site 2, Frankenberg
  - Boehringer Ingelheim Investigational Site 3, Frankenberg
  - Boehringer Ingelheim Investigational Site 10, Frankfurt
  - Boehringer Ingelheim Investigational Site 11, Frankfurt
  - Boehringer Ingelheim Investigational Site 12, Frankfurt
  - Boehringer Ingelheim Investigational Site 13, Frankfurt
  - Boehringer Ingelheim Investigational Site 14, Frankfurt
  - Boehringer Ingelheim Investigational Site 15, Frankfurt
  - Boehringer Ingelheim Investigational Site 16, Frankfurt
  - Boehringer Ingelheim Investigational Site 17, Frankfurt
  - Boehringer Ingelheim Investigational Site 18, Frankfurt
  - Boehringer Ingelheim Investigational Site 19, Frankfurt
  - Boehringer Ingelheim Investigational Site 1, Frankfurt
  - Boehringer Ingelheim Investigational Site 2, Frankfurt
  - Boehringer Ingelheim Investigational Site 3, Frankfurt
  - Boehringer Ingelheim Investigational Site 4, Frankfurt
  - Boehringer Ingelheim Investigational Site 5, Frankfurt
  - Boehringer Ingelheim Investigational Site 6, Frankfurt
  - Boehringer Ingelheim Investigational Site 7, Frankfurt
  - Boehringer Ingelheim Investigational Site 8, Frankfurt
  - Boehringer Ingelheim Investigational Site 9, Frankfurt
  - Boehringer Ingelheim Investigational Site, Franzburg
  - Boehringer Ingelheim Investigational Site, Frechen
  - Boehringer Ingelheim Investigational Site 1, Freiberg
  - Boehringer Ingelheim Investigational Site 2, Freiberg
  - Boehringer Ingelheim Investigational Site 1, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 2, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 3, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 4, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 5, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 6, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site, Freilassing
  - Boehringer Ingelheim Investigational Site, Freinsheim
  - Boehringer Ingelheim Investigational Site 1, Freisen
  - Boehringer Ingelheim Investigational Site 2, Freisen
  - Boehringer Ingelheim Investigational Site, Freital
  - Boehringer Ingelheim Investigational Site 1, Freyung
  - Boehringer Ingelheim Investigational Site 2, Freyung
  - Boehringer Ingelheim Investigational Site, Friedberg
  - Boehringer Ingelheim Investigational Site 1, Friedrichshafen
  - Boehringer Ingelheim Investigational Site 2, Friedrichshafen
  - Boehringer Ingelheim Investigational Site 1, Friedrichsthal
  - Boehringer Ingelheim Investigational Site 2, Friedrichsthal
  - Boehringer Ingelheim Investigational Site 3, Friedrichsthal
  - Boehringer Ingelheim Investigational Site 4, Friedrichsthal
  - Boehringer Ingelheim Investigational Site 5, Friedrichsthal
  - Boehringer Ingelheim Investigational Site 1, Friesoythe
  - Boehringer Ingelheim Investigational Site 2, Friesoythe
  - Boehringer Ingelheim Investigational Site, Friolzheim
  - Boehringer Ingelheim Investigational Site, Frohburg
  - Boehringer Ingelheim Investigational Site, Fuchsstadt
  - Boehringer Ingelheim Investigational Site, Fulda
  - Boehringer Ingelheim Investigational Site, Furth im Wald
  - Boehringer Ingelheim Investigational Site, Fußgönheim
  - Boehringer Ingelheim Investigational Site, Fürstenzell
  - Boehringer Ingelheim Investigational Site 1, Fürth
  - Boehringer Ingelheim Investigational Site 2, Fürth
  - Boehringer Ingelheim Investigational Site 3, Fürth
  - Boehringer Ingelheim Investigational Site 4, Fürth
  - Boehringer Ingelheim Investigational Site, Gaggenau
  - Boehringer Ingelheim Investigational Site, Gaildorf
  - Boehringer Ingelheim Investigational Site, Ganderkesee
  - Boehringer Ingelheim Investigational Site 1, Gangelt
  - Boehringer Ingelheim Investigational Site 2, Gangelt
  - Boehringer Ingelheim Investigational Site 1, Garbsen
  - Boehringer Ingelheim Investigational Site 2, Garbsen
  - Boehringer Ingelheim Investigational Site, Garching
  - Boehringer Ingelheim Investigational Site, Garmisch-Partenkirchen
  - Boehringer Ingelheim Investigational Site, Gau-Bischofsheim
  - Boehringer Ingelheim Investigational Site, Gechingen
  - Boehringer Ingelheim Investigational Site, Gefrees
  - Boehringer Ingelheim Investigational Site, Geisenheim
  - Boehringer Ingelheim Investigational Site 1, Gelnhausen
  - Boehringer Ingelheim Investigational Site 2, Gelnhausen
  - Boehringer Ingelheim Investigational Site 3, Gelnhausen
  - Boehringer Ingelheim Investigational Site 10, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 11, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 12, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 1, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 2, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 3, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 4, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 5, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 6, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 7, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 8, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 9, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site, Gengenbach
  - Boehringer Ingelheim Investigational Site, Gensingen
  - Boehringer Ingelheim Investigational Site, Genthin
  - Boehringer Ingelheim Investigational Site, Georgsmarienhütte
  - Boehringer Ingelheim Investigational Site 1, Gera
  - Boehringer Ingelheim Investigational Site 2, Gera
  - Boehringer Ingelheim Investigational Site 3, Gera
  - Boehringer Ingelheim Investigational Site 4, Gera
  - Boehringer Ingelheim Investigational Site 5, Gera
  - Boehringer Ingelheim Investigational Site 6, Gera
  - Boehringer Ingelheim Investigational Site 7, Gera
  - Boehringer Ingelheim Investigational Site 1, Geretsried
  - Boehringer Ingelheim Investigational Site 2, Geretsried
  - Boehringer Ingelheim Investigational Site, Germering
  - Boehringer Ingelheim Investigational Site, Germersheim
  - Boehringer Ingelheim Investigational Site, Gersfeld
  - Boehringer Ingelheim Investigational Site, Gersthofen
  - Boehringer Ingelheim Investigational Site 1, Giessen
  - Boehringer Ingelheim Investigational Site 2, Giessen
  - Boehringer Ingelheim Investigational Site 3, Giessen
  - Boehringer Ingelheim Investigational Site 4, Giessen
  - Boehringer Ingelheim Investigational Site 5, Giessen
  - Boehringer Ingelheim Investigational Site, Gifhorn
  - Boehringer Ingelheim Investigational Site, Ginsheim-Gustavsburg
  - Boehringer Ingelheim Investigational Site 1, Gladbeck
  - Boehringer Ingelheim Investigational Site 2, Gladbeck
  - Boehringer Ingelheim Investigational Site 3, Gladbeck
  - Boehringer Ingelheim Investigational Site 4, Gladbeck
  - Boehringer Ingelheim Investigational Site 5, Gladbeck
  - Boehringer Ingelheim Investigational Site 6, Gladbeck
  - Boehringer Ingelheim Investigational Site, Glan-Münchweiler
  - Boehringer Ingelheim Investigational Site, Glashütten
  - Boehringer Ingelheim Investigational Site 1, Gleichen
  - Boehringer Ingelheim Investigational Site 2, Gleichen
  - Boehringer Ingelheim Investigational Site, Glienicke
  - Boehringer Ingelheim Investigational Site, Glücksburg
  - Boehringer Ingelheim Investigational Site, Goch
  - Boehringer Ingelheim Investigational Site, Gochsheim
  - Boehringer Ingelheim Investigational Site, Goldberg
  - Boehringer Ingelheim Investigational Site, Golzow
  - Boehringer Ingelheim Investigational Site, Gomaringen
  - Boehringer Ingelheim Investigational Site, Gommern
  - Boehringer Ingelheim Investigational Site, Görisried
  - Boehringer Ingelheim Investigational Site, Görlitz
  - Boehringer Ingelheim Investigational Site 1, Göttingen
  - Boehringer Ingelheim Investigational Site 2, Göttingen
  - Boehringer Ingelheim Investigational Site 3, Göttingen
  - Boehringer Ingelheim Investigational Site 4, Göttingen
  - Boehringer Ingelheim Investigational Site 5, Göttingen
  - Boehringer Ingelheim Investigational Site, Grafing
  - Boehringer Ingelheim Investigational Site, Gräfelfing
  - Boehringer Ingelheim Investigational Site, Gräfenhainichen
  - Boehringer Ingelheim Investigational Site, Gräfinau-Angstedt
  - Boehringer Ingelheim Investigational Site 1, Greiz
  - Boehringer Ingelheim Investigational Site 2, Greiz
  - Boehringer Ingelheim Investigational Site 1, Grevenbroich
  - Boehringer Ingelheim Investigational Site 2, Grevenbroich
  - Boehringer Ingelheim Investigational Site 3, Grevenbroich
  - Boehringer Ingelheim Investigational Site 4, Grevenbroich
  - Boehringer Ingelheim Investigational Site, Grimma
  - Boehringer Ingelheim Investigational Site, Groß Börnecke
  - Boehringer Ingelheim Investigational Site 1, Groß Leuthen
  - Boehringer Ingelheim Investigational Site 2, Groß Leuthen
  - Boehringer Ingelheim Investigational Site, Groß-Zimmern
  - Boehringer Ingelheim Investigational Site 1, Großefehn
  - Boehringer Ingelheim Investigational Site 2, Großefehn
  - Boehringer Ingelheim Investigational Site 3, Großefehn
  - Boehringer Ingelheim Investigational Site, Großen Buseck
  - Boehringer Ingelheim Investigational Site, Großenhain
  - Boehringer Ingelheim Investigational Site, Großenkneten
  - Boehringer Ingelheim Investigational Site, Großerkmannsdorf
  - Boehringer Ingelheim Investigational Site, Großerlach
  - Boehringer Ingelheim Investigational Site, Großfriesen
  - Boehringer Ingelheim Investigational Site, Großhabersdorf
  - Boehringer Ingelheim Investigational Site, Großkorbetha
  - Boehringer Ingelheim Investigational Site, Großkrotzenburg
  - Boehringer Ingelheim Investigational Site 1, Großmaischeid
  - Boehringer Ingelheim Investigational Site 2, Großmaischeid
  - Boehringer Ingelheim Investigational Site 1, Großräschen
  - Boehringer Ingelheim Investigational Site 2, Großräschen
  - Boehringer Ingelheim Investigational Site, Großrosseln
  - Boehringer Ingelheim Investigational Site, Großschirma
  - Boehringer Ingelheim Investigational Site, Grömitz
  - Boehringer Ingelheim Investigational Site, Grünheide
  - Boehringer Ingelheim Investigational Site, Gudensberg
  - Boehringer Ingelheim Investigational Site 1, Gummersbach
  - Boehringer Ingelheim Investigational Site 2, Gummersbach
  - Boehringer Ingelheim Investigational Site 3, Gummersbach
  - Boehringer Ingelheim Investigational Site 4, Gummersbach
  - Boehringer Ingelheim Investigational Site 5, Gummersbach
  - Boehringer Ingelheim Investigational Site, Gundheim
  - Boehringer Ingelheim Investigational Site, Guntersblum
  - Boehringer Ingelheim Investigational Site, Gunzenhausen
  - Boehringer Ingelheim Investigational Site 1, Guxhagen
  - Boehringer Ingelheim Investigational Site 2, Guxhagen
  - Boehringer Ingelheim Investigational Site, Güntersleben
  - Boehringer Ingelheim Investigational Site, Güstrow
  - Boehringer Ingelheim Investigational Site 1, Gütersloh
  - Boehringer Ingelheim Investigational Site 2, Gütersloh
  - Boehringer Ingelheim Investigational Site 3, Gütersloh
  - Boehringer Ingelheim Investigational Site 4, Gütersloh
  - Boehringer Ingelheim Investigational Site 1, Haag
  - Boehringer Ingelheim Investigational Site 2, Haag
  - Boehringer Ingelheim Investigational Site 1, Haar
  - Boehringer Ingelheim Investigational Site 2, Haar
  - Boehringer Ingelheim Investigational Site 1, Hagen
  - Boehringer Ingelheim Investigational Site 2, Hagen
  - Boehringer Ingelheim Investigational Site 3, Hagen
  - Boehringer Ingelheim Investigational Site 4, Hagen
  - Boehringer Ingelheim Investigational Site 5, Hagen
  - Boehringer Ingelheim Investigational Site 6, Hagen
  - Boehringer Ingelheim Investigational Site 7, Hagen
  - Boehringer Ingelheim Investigational Site 8, Hagen
  - Boehringer Ingelheim Investigational Site 9, Hagen
  - Boehringer Ingelheim Investigational Site 1, Hagenow
  - Boehringer Ingelheim Investigational Site 2, Hagenow
  - Boehringer Ingelheim Investigational Site, Haigerloch
  - Boehringer Ingelheim Investigational Site 1, Hainburg
  - Boehringer Ingelheim Investigational Site 2, Hainburg
  - Boehringer Ingelheim Investigational Site, Halbe
  - Boehringer Ingelheim Investigational Site 1, Haldensleben I
  - Boehringer Ingelheim Investigational Site 2, Haldensleben I
  - Boehringer Ingelheim Investigational Site 10, Halle
  - Boehringer Ingelheim Investigational Site 11, Halle
  - Boehringer Ingelheim Investigational Site 12, Halle
  - Boehringer Ingelheim Investigational Site 13, Halle
  - Boehringer Ingelheim Investigational Site 14, Halle
  - Boehringer Ingelheim Investigational Site 15, Halle
  - Boehringer Ingelheim Investigational Site 16, Halle
  - Boehringer Ingelheim Investigational Site 17, Halle
  - Boehringer Ingelheim Investigational Site 18, Halle
  - Boehringer Ingelheim Investigational Site 19, Halle
  - Boehringer Ingelheim Investigational Site 1, Halle
  - Boehringer Ingelheim Investigational Site 20, Halle
  - Boehringer Ingelheim Investigational Site 21, Halle
  - Boehringer Ingelheim Investigational Site 22, Halle
  - Boehringer Ingelheim Investigational Site 2, Halle
  - Boehringer Ingelheim Investigational Site 3, Halle
  - Boehringer Ingelheim Investigational Site 4, Halle
  - Boehringer Ingelheim Investigational Site 5, Halle
  - Boehringer Ingelheim Investigational Site 6, Halle
  - Boehringer Ingelheim Investigational Site 7, Halle
  - Boehringer Ingelheim Investigational Site 8, Halle
  - Boehringer Ingelheim Investigational Site 9, Halle
  - Boehringer Ingelheim Investigational Site, Hallstadt
  - Boehringer Ingelheim Investigational Site, Halver
  - Boehringer Ingelheim Investigational Site 10, Hamburg
  - Boehringer Ingelheim Investigational Site 11, Hamburg
  - Boehringer Ingelheim Investigational Site 12, Hamburg
  - Boehringer Ingelheim Investigational Site 13, Hamburg
  - Boehringer Ingelheim Investigational Site 14, Hamburg
  - Boehringer Ingelheim Investigational Site 15, Hamburg
  - Boehringer Ingelheim Investigational Site 16, Hamburg
  - Boehringer Ingelheim Investigational Site 17, Hamburg
  - Boehringer Ingelheim Investigational Site 18, Hamburg
  - Boehringer Ingelheim Investigational Site 19, Hamburg
  - Boehringer Ingelheim Investigational Site 1, Hamburg
  - Boehringer Ingelheim Investigational Site 20, Hamburg
  - Boehringer Ingelheim Investigational Site 21, Hamburg
  - Boehringer Ingelheim Investigational Site 22, Hamburg
  - Boehringer Ingelheim Investigational Site 23, Hamburg
  - Boehringer Ingelheim Investigational Site 24, Hamburg
  - Boehringer Ingelheim Investigational Site 25, Hamburg
  - Boehringer Ingelheim Investigational Site 26, Hamburg
  - Boehringer Ingelheim Investigational Site 27, Hamburg
  - Boehringer Ingelheim Investigational Site 28, Hamburg
  - Boehringer Ingelheim Investigational Site 29, Hamburg
  - Boehringer Ingelheim Investigational Site 2, Hamburg
  - Boehringer Ingelheim Investigational Site 30, Hamburg
  - Boehringer Ingelheim Investigational Site 31, Hamburg
  - Boehringer Ingelheim Investigational Site 32, Hamburg
  - Boehringer Ingelheim Investigational Site 33, Hamburg
  - Boehringer Ingelheim Investigational Site 34, Hamburg
  - Boehringer Ingelheim Investigational Site 35, Hamburg
  - Boehringer Ingelheim Investigational Site 36, Hamburg
  - Boehringer Ingelheim Investigational Site 37, Hamburg
  - Boehringer Ingelheim Investigational Site 38, Hamburg
  - Boehringer Ingelheim Investigational Site 39, Hamburg
  - Boehringer Ingelheim Investigational Site 3, Hamburg
  - Boehringer Ingelheim Investigational Site 40, Hamburg
  - Boehringer Ingelheim Investigational Site 41, Hamburg
  - Boehringer Ingelheim Investigational Site 42, Hamburg
  - Boehringer Ingelheim Investigational Site 4, Hamburg
  - Boehringer Ingelheim Investigational Site 5, Hamburg
  - Boehringer Ingelheim Investigational Site 6, Hamburg
  - Boehringer Ingelheim Investigational Site 7, Hamburg
  - Boehringer Ingelheim Investigational Site 8, Hamburg
  - Boehringer Ingelheim Investigational Site 9, Hamburg
  - Boehringer Ingelheim Investigational Site 1, Hamelin
  - Boehringer Ingelheim Investigational Site 2, Hamelin
  - Boehringer Ingelheim Investigational Site 10, Hamm
  - Boehringer Ingelheim Investigational Site 1, Hamm
  - Boehringer Ingelheim Investigational Site 2, Hamm
  - Boehringer Ingelheim Investigational Site 3, Hamm
  - Boehringer Ingelheim Investigational Site 4, Hamm
  - Boehringer Ingelheim Investigational Site 5, Hamm
  - Boehringer Ingelheim Investigational Site 6, Hamm
  - Boehringer Ingelheim Investigational Site 7, Hamm
  - Boehringer Ingelheim Investigational Site 8, Hamm
  - Boehringer Ingelheim Investigational Site 9, Hamm
  - Boehringer Ingelheim Investigational Site, Hammah
  - Boehringer Ingelheim Investigational Site, Hammelburg
  - Boehringer Ingelheim Investigational Site, Hamminkeln
  - Boehringer Ingelheim Investigational Site 1, Hanau
  - Boehringer Ingelheim Investigational Site 2, Hanau
  - Boehringer Ingelheim Investigational Site 3, Hanau
  - Boehringer Ingelheim Investigational Site 4, Hanau
  - Boehringer Ingelheim Investigational Site 5, Hanau
  - Boehringer Ingelheim Investigational Site 10, Hanover
  - Boehringer Ingelheim Investigational Site 11, Hanover
  - Boehringer Ingelheim Investigational Site 12, Hanover
  - Boehringer Ingelheim Investigational Site 13, Hanover
  - Boehringer Ingelheim Investigational Site 1, Hanover
  - Boehringer Ingelheim Investigational Site 2, Hanover
  - Boehringer Ingelheim Investigational Site 3, Hanover
  - Boehringer Ingelheim Investigational Site 4, Hanover
  - Boehringer Ingelheim Investigational Site 5, Hanover
  - Boehringer Ingelheim Investigational Site 6, Hanover
  - Boehringer Ingelheim Investigational Site 7, Hanover
  - Boehringer Ingelheim Investigational Site 8, Hanover
  - Boehringer Ingelheim Investigational Site 9, Hanover
  - Boehringer Ingelheim Investigational Site, Haren
  - Boehringer Ingelheim Investigational Site 1, Harsewinkel
  - Boehringer Ingelheim Investigational Site 2, Harsewinkel
  - Boehringer Ingelheim Investigational Site 3, Harsewinkel
  - Boehringer Ingelheim Investigational Site, Hartenstein
  - Boehringer Ingelheim Investigational Site, Harzgerode
  - Boehringer Ingelheim Investigational Site, Haselbachtal
  - Boehringer Ingelheim Investigational Site, Haselünne
  - Boehringer Ingelheim Investigational Site, Hatten
  - Boehringer Ingelheim Investigational Site, Hattingen
  - Boehringer Ingelheim Investigational Site, Hattorf
  - Boehringer Ingelheim Investigational Site, Haunsheim
  - Boehringer Ingelheim Investigational Site, Haßloch
  - Boehringer Ingelheim Investigational Site, Heddesheim
  - Boehringer Ingelheim Investigational Site 1, Heek
  - Boehringer Ingelheim Investigational Site 2, Heek
  - Boehringer Ingelheim Investigational Site 3, Heek
  - Boehringer Ingelheim Investigational Site, Heeslingen
  - Boehringer Ingelheim Investigational Site 1, Heidelberg
  - Boehringer Ingelheim Investigational Site 2, Heidelberg
  - Boehringer Ingelheim Investigational Site 3, Heidelberg
  - Boehringer Ingelheim Investigational Site 4, Heidelberg
  - Boehringer Ingelheim Investigational Site, Heidenheim
  - Boehringer Ingelheim Investigational Site, Heilbad Heiligenstadt
  - Boehringer Ingelheim Investigational Site 1, Heilbronn
  - Boehringer Ingelheim Investigational Site 2, Heilbronn
  - Boehringer Ingelheim Investigational Site 3, Heilbronn
  - Boehringer Ingelheim Investigational Site, Heiligenhafen
  - Boehringer Ingelheim Investigational Site, Heilsbronn
  - Boehringer Ingelheim Investigational Site 1, Heimsheim
  - Boehringer Ingelheim Investigational Site 2, Heimsheim
  - Boehringer Ingelheim Investigational Site 1, Heinsberg
  - Boehringer Ingelheim Investigational Site 2, Heinsberg
  - Boehringer Ingelheim Investigational Site, Hellenthal
  - Boehringer Ingelheim Investigational Site 1, Helmstedt
  - Boehringer Ingelheim Investigational Site 2, Helmstedt
  - Boehringer Ingelheim Investigational Site 1, Hemer
  - Boehringer Ingelheim Investigational Site 2, Hemer
  - Boehringer Ingelheim Investigational Site 3, Hemer
  - Boehringer Ingelheim Investigational Site, Hennigsdorf
  - Boehringer Ingelheim Investigational Site, Henstedt-Ulzburg
  - Boehringer Ingelheim Investigational Site, Heppenheim an der Bergstrasse
  - Boehringer Ingelheim Investigational Site, Herborn
  - Boehringer Ingelheim Investigational Site, Herbsleben
  - Boehringer Ingelheim Investigational Site, Herdecke
  - Boehringer Ingelheim Investigational Site, Herford
  - Boehringer Ingelheim Investigational Site, Heringen
  - Boehringer Ingelheim Investigational Site 1, Herne
  - Boehringer Ingelheim Investigational Site 2, Herne
  - Boehringer Ingelheim Investigational Site 3, Herne
  - Boehringer Ingelheim Investigational Site 4, Herne
  - Boehringer Ingelheim Investigational Site 5, Herne
  - Boehringer Ingelheim Investigational Site, Herrenberg
  - Boehringer Ingelheim Investigational Site, Herrnhut
  - Boehringer Ingelheim Investigational Site, Herscheid
  - Boehringer Ingelheim Investigational Site, Herzogenaurach
  - Boehringer Ingelheim Investigational Site, Hesel
  - Boehringer Ingelheim Investigational Site, Hessisch Lichtenau
  - Boehringer Ingelheim Investigational Site, Hessisch Oldendorf
  - Boehringer Ingelheim Investigational Site, Hettstedt
  - Boehringer Ingelheim Investigational Site, Hetzerath
  - Boehringer Ingelheim Investigational Site, Heßdorf
  - Boehringer Ingelheim Investigational Site 1, Hiddenhausen
  - Boehringer Ingelheim Investigational Site 2, Hiddenhausen
  - Boehringer Ingelheim Investigational Site, Hilders
  - Boehringer Ingelheim Investigational Site 1, Hildesheim
  - Boehringer Ingelheim Investigational Site 2, Hildesheim
  - Boehringer Ingelheim Investigational Site, Hillersleben
  - Boehringer Ingelheim Investigational Site, Hinterhermsdorf
  - Boehringer Ingelheim Investigational Site, Hirschaid
  - Boehringer Ingelheim Investigational Site, Hof
  - Boehringer Ingelheim Investigational Site 1, Hofheim
  - Boehringer Ingelheim Investigational Site 2, Hofheim
  - Boehringer Ingelheim Investigational Site, Hohen Neuendorf
  - Boehringer Ingelheim Investigational Site, Hohenpeißenberg
  - Boehringer Ingelheim Investigational Site, Hohenwart
  - Boehringer Ingelheim Investigational Site, Hollfeld
  - Boehringer Ingelheim Investigational Site, Homburg
  - Boehringer Ingelheim Investigational Site, Horb
  - Boehringer Ingelheim Investigational Site, Horn-Bad Meinberg
  - Boehringer Ingelheim Investigational Site 1, Hoyerswerda
  - Boehringer Ingelheim Investigational Site 2, Hoyerswerda
  - Boehringer Ingelheim Investigational Site 3, Hoyerswerda
  - Boehringer Ingelheim Investigational Site 4, Hoyerswerda
  - Boehringer Ingelheim Investigational Site, Hoym
  - Boehringer Ingelheim Investigational Site, Höchheim
  - Boehringer Ingelheim Investigational Site, Höhn
  - Boehringer Ingelheim Investigational Site, Hörstel
  - Boehringer Ingelheim Investigational Site, Hösbach
  - Boehringer Ingelheim Investigational Site, Hötensleben
  - Boehringer Ingelheim Investigational Site, Hundshübel
  - Boehringer Ingelheim Investigational Site, Husby
  - Boehringer Ingelheim Investigational Site, Huska
  - Boehringer Ingelheim Investigational Site 1, Hückeswagen
  - Boehringer Ingelheim Investigational Site 2, Hückeswagen
  - Boehringer Ingelheim Investigational Site 1, Hüllhorst
  - Boehringer Ingelheim Investigational Site 2, Hüllhorst
  - Boehringer Ingelheim Investigational Site, Hünfelden
  - Boehringer Ingelheim Investigational Site, Ifta
  - Boehringer Ingelheim Investigational Site, Ihlienworth
  - Boehringer Ingelheim Investigational Site 1, Illingen
  - Boehringer Ingelheim Investigational Site 2, Illingen
  - Boehringer Ingelheim Investigational Site 1, Ilmenau
  - Boehringer Ingelheim Investigational Site 2, Ilmenau
  - Boehringer Ingelheim Investigational Site 3, Ilmenau
  - Boehringer Ingelheim Investigational Site, Ilsede
  - Boehringer Ingelheim Investigational Site, Ilsfeld
  - Boehringer Ingelheim Investigational Site, Ingelheim
  - Boehringer Ingelheim Investigational Site, Ingersheim
  - Boehringer Ingelheim Investigational Site 1, Ingolstadt
  - Boehringer Ingelheim Investigational Site 2, Ingolstadt
  - Boehringer Ingelheim Investigational Site 1, Iserlohn
  - Boehringer Ingelheim Investigational Site 2, Iserlohn
  - Boehringer Ingelheim Investigational Site 3, Iserlohn
  - Boehringer Ingelheim Investigational Site 4, Iserlohn
  - Boehringer Ingelheim Investigational Site 5, Iserlohn
  - Boehringer Ingelheim Investigational Site 1, Isernhagen-Süd
  - Boehringer Ingelheim Investigational Site 2, Isernhagen-Süd
  - Boehringer Ingelheim Investigational Site, Issum
  - Boehringer Ingelheim Investigational Site, Jahnsdorf
  - Boehringer Ingelheim Investigational Site 1, Jena
  - Boehringer Ingelheim Investigational Site 2, Jena
  - Boehringer Ingelheim Investigational Site 3, Jena
  - Boehringer Ingelheim Investigational Site 4, Jena
  - Boehringer Ingelheim Investigational Site, Jerxheim
  - Boehringer Ingelheim Investigational Site, Jettingen
  - Boehringer Ingelheim Investigational Site, Johannesberg
  - Boehringer Ingelheim Investigational Site 1, Jübek
  - Boehringer Ingelheim Investigational Site 2, Jübek
  - Boehringer Ingelheim Investigational Site, Jühnde
  - Boehringer Ingelheim Investigational Site 1, Jüterbog
  - Boehringer Ingelheim Investigational Site 2, Jüterbog
  - Boehringer Ingelheim Investigational Site, Kaarst
  - Boehringer Ingelheim Investigational Site 1, Kaiserslautern
  - Boehringer Ingelheim Investigational Site 2, Kaiserslautern
  - Boehringer Ingelheim Investigational Site, Kalawa
  - Boehringer Ingelheim Investigational Site, Kalkar
  - Boehringer Ingelheim Investigational Site, Kalkhorst
  - Boehringer Ingelheim Investigational Site, Kall
  - Boehringer Ingelheim Investigational Site, Kamen
  - Boehringer Ingelheim Investigational Site, Kamenz
  - Boehringer Ingelheim Investigational Site, Kammerforst
  - Boehringer Ingelheim Investigational Site, Kamp-Bornhofen
  - Boehringer Ingelheim Investigational Site, Kamp-Lintfort
  - Boehringer Ingelheim Investigational Site, Kappeln
  - Boehringer Ingelheim Investigational Site, Kappelrodeck
  - Boehringer Ingelheim Investigational Site, Karlskron
  - Boehringer Ingelheim Investigational Site 1, Karlsruhe
  - Boehringer Ingelheim Investigational Site 2, Karlsruhe
  - Boehringer Ingelheim Investigational Site 3, Karlsruhe
  - Boehringer Ingelheim Investigational Site 4, Karlsruhe
  - Boehringer Ingelheim Investigational Site, Karlstadt am Main
  - Boehringer Ingelheim Investigational Site 10, Kassel
  - Boehringer Ingelheim Investigational Site 11, Kassel
  - Boehringer Ingelheim Investigational Site 1, Kassel
  - Boehringer Ingelheim Investigational Site 2, Kassel
  - Boehringer Ingelheim Investigational Site 3, Kassel
  - Boehringer Ingelheim Investigational Site 4, Kassel
  - Boehringer Ingelheim Investigational Site 5, Kassel
  - Boehringer Ingelheim Investigational Site 6, Kassel
  - Boehringer Ingelheim Investigational Site 7, Kassel
  - Boehringer Ingelheim Investigational Site 8, Kassel
  - Boehringer Ingelheim Investigational Site 9, Kassel
  - Boehringer Ingelheim Investigational Site, Katlenburg-Lindau
  - Boehringer Ingelheim Investigational Site, Katzenelnbogen
  - Boehringer Ingelheim Investigational Site 1, Katzhütte
  - Boehringer Ingelheim Investigational Site 2, Katzhütte
  - Boehringer Ingelheim Investigational Site 1, Kaufbeuren
  - Boehringer Ingelheim Investigational Site 2, Kaufbeuren
  - Boehringer Ingelheim Investigational Site 3, Kaufbeuren
  - Boehringer Ingelheim Investigational Site 4, Kaufbeuren
  - Boehringer Ingelheim Investigational Site, Keltern
  - Boehringer Ingelheim Investigational Site 1, Kempen
  - Boehringer Ingelheim Investigational Site 2, Kempen
  - Boehringer Ingelheim Investigational Site 3, Kempen
  - Boehringer Ingelheim Investigational Site, Kempenich
  - Boehringer Ingelheim Investigational Site 1, Kempten
  - Boehringer Ingelheim Investigational Site 2, Kempten
  - Boehringer Ingelheim Investigational Site 3, Kempten
  - Boehringer Ingelheim Investigational Site, Kenzingen
  - Boehringer Ingelheim Investigational Site, Kernen
  - Boehringer Ingelheim Investigational Site 1, Kerpen
  - Boehringer Ingelheim Investigational Site 2, Kerpen
  - Boehringer Ingelheim Investigational Site, Kiedrich
  - Boehringer Ingelheim Investigational Site 1, Kiel
  - Boehringer Ingelheim Investigational Site 2, Kiel
  - Boehringer Ingelheim Investigational Site, Kindsbach
  - Boehringer Ingelheim Investigational Site, Kippenheim
  - Boehringer Ingelheim Investigational Site, Kirchberg I. Wald
  - Boehringer Ingelheim Investigational Site, Kirchenlamitz
  - Boehringer Ingelheim Investigational Site 1, Kirchhain
  - Boehringer Ingelheim Investigational Site 2, Kirchhain
  - Boehringer Ingelheim Investigational Site 3, Kirchhain
  - Boehringer Ingelheim Investigational Site, Kirchhain
  - Boehringer Ingelheim Investigational Site, Kirchheimbolanden
  - Boehringer Ingelheim Investigational Site, Kirchhundem
  - Boehringer Ingelheim Investigational Site, Kirchlengern
  - Boehringer Ingelheim Investigational Site, Kirkel
  - Boehringer Ingelheim Investigational Site, Klausdorf
  - Boehringer Ingelheim Investigational Site 1, Kleinmachnow
  - Boehringer Ingelheim Investigational Site 2, Kleinmachnow
  - Boehringer Ingelheim Investigational Site 1, Kleve
  - Boehringer Ingelheim Investigational Site 2, Kleve
  - Boehringer Ingelheim Investigational Site, Klingenberg
  - Boehringer Ingelheim Investigational Site, Kloster Lehnin
  - Boehringer Ingelheim Investigational Site 1, Koblenz
  - Boehringer Ingelheim Investigational Site 2, Koblenz
  - Boehringer Ingelheim Investigational Site 3, Koblenz
  - Boehringer Ingelheim Investigational Site 4, Koblenz
  - Boehringer Ingelheim Investigational Site, Kolitzheim
  - Boehringer Ingelheim Investigational Site, Konstanz
  - Boehringer Ingelheim Investigational Site, Kornwestheim
  - Boehringer Ingelheim Investigational Site, Koßdorf
  - Boehringer Ingelheim Investigational Site, Königerode
  - Boehringer Ingelheim Investigational Site, Königs Wusterhausen
  - Boehringer Ingelheim Investigational Site, Königsberg
  - Boehringer Ingelheim Investigational Site, Königsbrück
  - Boehringer Ingelheim Investigational Site, Kösching
  - Boehringer Ingelheim Investigational Site 1, Köthen
  - Boehringer Ingelheim Investigational Site 2, Köthen
  - Boehringer Ingelheim Investigational Site 3, Köthen
  - Boehringer Ingelheim Investigational Site 1, Krefeld
  - Boehringer Ingelheim Investigational Site 2, Krefeld
  - Boehringer Ingelheim Investigational Site 3, Krefeld
  - Boehringer Ingelheim Investigational Site 4, Krefeld
  - Boehringer Ingelheim Investigational Site 5, Krefeld
  - Boehringer Ingelheim Investigational Site 6, Krefeld
  - Boehringer Ingelheim Investigational Site 7, Krefeld
  - Boehringer Ingelheim Investigational Site 8, Krefeld
  - Boehringer Ingelheim Investigational Site, Kressbronn
  - Boehringer Ingelheim Investigational Site 1, Kreuztal
  - Boehringer Ingelheim Investigational Site 2, Kreuztal
  - Boehringer Ingelheim Investigational Site 1, Kronach
  - Boehringer Ingelheim Investigational Site 2, Kronach
  - Boehringer Ingelheim Investigational Site, Kronberg
  - Boehringer Ingelheim Investigational Site, Kronshagen
  - Boehringer Ingelheim Investigational Site, Krumbach
  - Boehringer Ingelheim Investigational Site, Krummennaab
  - Boehringer Ingelheim Investigational Site, Kuchen
  - Boehringer Ingelheim Investigational Site, Kulmbach
  - Boehringer Ingelheim Investigational Site, Kupferzell
  - Boehringer Ingelheim Investigational Site 1, Kusel
  - Boehringer Ingelheim Investigational Site 2, Kusel
  - Boehringer Ingelheim Investigational Site, Kümmersbruck
  - Boehringer Ingelheim Investigational Site, Künzell
  - Boehringer Ingelheim Investigational Site 1, Künzelsau
  - Boehringer Ingelheim Investigational Site 2, Künzelsau
  - Boehringer Ingelheim Investigational Site, Künzing
  - Boehringer Ingelheim Investigational Site, Küps
  - Boehringer Ingelheim Investigational Site 1, Laatzen
  - Boehringer Ingelheim Investigational Site 2, Laatzen
  - Boehringer Ingelheim Investigational Site 3, Laatzen
  - Boehringer Ingelheim Investigational Site 1, Lahnau
  - Boehringer Ingelheim Investigational Site 2, Lahnau
  - Boehringer Ingelheim Investigational Site, Lahntal
  - Boehringer Ingelheim Investigational Site, Lahr
  - Boehringer Ingelheim Investigational Site, Lalendorf
  - Boehringer Ingelheim Investigational Site, Lalling
  - Boehringer Ingelheim Investigational Site, Landau
  - Boehringer Ingelheim Investigational Site, Landsberg
  - Boehringer Ingelheim Investigational Site, Landshut
  - Boehringer Ingelheim Investigational Site, Landstuhl
  - Boehringer Ingelheim Investigational Site, Langen
  - Boehringer Ingelheim Investigational Site, Langenbogen
  - Boehringer Ingelheim Investigational Site, Langenenslingen
  - Boehringer Ingelheim Investigational Site 1, Langenfeld
  - Boehringer Ingelheim Investigational Site 2, Langenfeld
  - Boehringer Ingelheim Investigational Site 3, Langenfeld
  - Boehringer Ingelheim Investigational Site 4, Langenfeld
  - Boehringer Ingelheim Investigational Site, Langenzenn
  - Boehringer Ingelheim Investigational Site, Langweid
  - Boehringer Ingelheim Investigational Site, Lassan
  - Boehringer Ingelheim Investigational Site, Lastrup
  - Boehringer Ingelheim Investigational Site, Laubusch
  - Boehringer Ingelheim Investigational Site, Lauchringen
  - Boehringer Ingelheim Investigational Site, Lauf
  - Boehringer Ingelheim Investigational Site, Lauffen am Neckar
  - Boehringer Ingelheim Investigational Site, Lauterecken
  - Boehringer Ingelheim Investigational Site, Lebach
  - Boehringer Ingelheim Investigational Site, Leck
  - Boehringer Ingelheim Investigational Site 1, Leer
  - Boehringer Ingelheim Investigational Site 2, Leer
  - Boehringer Ingelheim Investigational Site 3, Leer
  - Boehringer Ingelheim Investigational Site, Leezen
  - Boehringer Ingelheim Investigational Site, Legden
  - Boehringer Ingelheim Investigational Site, Leimen
  - Boehringer Ingelheim Investigational Site, Leimersheim
  - Boehringer Ingelheim Investigational Site, Leipheim
  - Boehringer Ingelheim Investigational Site 10, Leipzig
  - Boehringer Ingelheim Investigational Site 11, Leipzig
  - Boehringer Ingelheim Investigational Site 12, Leipzig
  - Boehringer Ingelheim Investigational Site 13, Leipzig
  - Boehringer Ingelheim Investigational Site 14, Leipzig
  - Boehringer Ingelheim Investigational Site 15, Leipzig
  - Boehringer Ingelheim Investigational Site 16, Leipzig
  - Boehringer Ingelheim Investigational Site 17, Leipzig
  - Boehringer Ingelheim Investigational Site 18, Leipzig
  - Boehringer Ingelheim Investigational Site 19, Leipzig
  - Boehringer Ingelheim Investigational Site 1, Leipzig
  - Boehringer Ingelheim Investigational Site 20, Leipzig
  - Boehringer Ingelheim Investigational Site 21, Leipzig
  - Boehringer Ingelheim Investigational Site 22, Leipzig
  - Boehringer Ingelheim Investigational Site 23, Leipzig
  - Boehringer Ingelheim Investigational Site 24, Leipzig
  - Boehringer Ingelheim Investigational Site 25, Leipzig
  - Boehringer Ingelheim Investigational Site 26, Leipzig
  - Boehringer Ingelheim Investigational Site 2, Leipzig
  - Boehringer Ingelheim Investigational Site 3, Leipzig
  - Boehringer Ingelheim Investigational Site 4, Leipzig
  - Boehringer Ingelheim Investigational Site 5, Leipzig
  - Boehringer Ingelheim Investigational Site 6, Leipzig
  - Boehringer Ingelheim Investigational Site 7, Leipzig
  - Boehringer Ingelheim Investigational Site 8, Leipzig
  - Boehringer Ingelheim Investigational Site 9, Leipzig
  - Boehringer Ingelheim Investigational Site 1, Lemförde
  - Boehringer Ingelheim Investigational Site 2, Lemförde
  - Boehringer Ingelheim Investigational Site, Lemgo
  - Boehringer Ingelheim Investigational Site, Leukersdorf
  - Boehringer Ingelheim Investigational Site, Leutenbach
  - Boehringer Ingelheim Investigational Site, Leutershausen
  - Boehringer Ingelheim Investigational Site 1, Leverkusen
  - Boehringer Ingelheim Investigational Site 2, Leverkusen
  - Boehringer Ingelheim Investigational Site 3, Leverkusen
  - Boehringer Ingelheim Investigational Site 4, Leverkusen
  - Boehringer Ingelheim Investigational Site 5, Leverkusen
  - Boehringer Ingelheim Investigational Site 6, Leverkusen
  - Boehringer Ingelheim Investigational Site, Lichtenfels
  - Boehringer Ingelheim Investigational Site, Liebenau
  - Boehringer Ingelheim Investigational Site 1, Lienen
  - Boehringer Ingelheim Investigational Site 2, Lienen
  - Boehringer Ingelheim Investigational Site, Limbach
  - Boehringer Ingelheim Investigational Site, Limburgerhof
  - Boehringer Ingelheim Investigational Site, Lindern
  - Boehringer Ingelheim Investigational Site 1, Linnich
  - Boehringer Ingelheim Investigational Site 2, Linnich
  - Boehringer Ingelheim Investigational Site, Linsengericht
  - Boehringer Ingelheim Investigational Site, Linz
  - Boehringer Ingelheim Investigational Site, Lippetal
  - Boehringer Ingelheim Investigational Site 1, Lippstadt
  - Boehringer Ingelheim Investigational Site 2, Lippstadt
  - Boehringer Ingelheim Investigational Site 3, Lippstadt
  - Boehringer Ingelheim Investigational Site 4, Lippstadt
  - Boehringer Ingelheim Investigational Site, Loerrach
  - Boehringer Ingelheim Investigational Site, Lohfelden
  - Boehringer Ingelheim Investigational Site, Lohmar
  - Boehringer Ingelheim Investigational Site, Lohsa
  - Boehringer Ingelheim Investigational Site 1, Lollar
  - Boehringer Ingelheim Investigational Site 2, Lollar
  - Boehringer Ingelheim Investigational Site, Losheim
  - Boehringer Ingelheim Investigational Site, Lotte
  - Boehringer Ingelheim Investigational Site, Löderburg
  - Boehringer Ingelheim Investigational Site 1, Löhne
  - Boehringer Ingelheim Investigational Site 2, Löhne
  - Boehringer Ingelheim Investigational Site 1, Lubnjow
  - Boehringer Ingelheim Investigational Site 2, Lubnjow
  - Boehringer Ingelheim Investigational Site 3, Lubnjow
  - Boehringer Ingelheim Investigational Site 4, Lubnjow
  - Boehringer Ingelheim Investigational Site 5, Lubnjow
  - Boehringer Ingelheim Investigational Site, Luckenwalde
  - Boehringer Ingelheim Investigational Site 1, Ludwigshafen
  - Boehringer Ingelheim Investigational Site 2, Ludwigshafen
  - Boehringer Ingelheim Investigational Site 3, Ludwigshafen
  - Boehringer Ingelheim Investigational Site 4, Ludwigshafen
  - Boehringer Ingelheim Investigational Site 5, Ludwigshafen
  - Boehringer Ingelheim Investigational Site 6, Ludwigshafen
  - Boehringer Ingelheim Investigational Site, Ludwigsstadt
  - Boehringer Ingelheim Investigational Site, Lutzerath
  - Boehringer Ingelheim Investigational Site 1, Lübbecke
  - Boehringer Ingelheim Investigational Site 2, Lübbecke
  - Boehringer Ingelheim Investigational Site 1, Lübeck
  - Boehringer Ingelheim Investigational Site 2, Lübeck
  - Boehringer Ingelheim Investigational Site 3, Lübeck
  - Boehringer Ingelheim Investigational Site 4, Lübeck
  - Boehringer Ingelheim Investigational Site 5, Lübeck
  - Boehringer Ingelheim Investigational Site 1, Lüdenscheid
  - Boehringer Ingelheim Investigational Site 2, Lüdenscheid
  - Boehringer Ingelheim Investigational Site 3, Lüdenscheid
  - Boehringer Ingelheim Investigational Site 4, Lüdenscheid
  - Boehringer Ingelheim Investigational Site 5, Lüdenscheid
  - Boehringer Ingelheim Investigational Site, Lügde
  - Boehringer Ingelheim Investigational Site, Lühmannsdorf
  - Boehringer Ingelheim Investigational Site 1, Lüneburg
  - Boehringer Ingelheim Investigational Site 2, Lüneburg
  - Boehringer Ingelheim Investigational Site 1, Lünen
  - Boehringer Ingelheim Investigational Site 2, Lünen
  - Boehringer Ingelheim Investigational Site 3, Lünen
  - Boehringer Ingelheim Investigational Site 4, Lünen
  - Boehringer Ingelheim Investigational Site 5, Lünen
  - Boehringer Ingelheim Investigational Site 6, Lünen
  - Boehringer Ingelheim Investigational Site 10, Magdeburg
  - Boehringer Ingelheim Investigational Site 11, Magdeburg
  - Boehringer Ingelheim Investigational Site 12, Magdeburg
  - Boehringer Ingelheim Investigational Site 13, Magdeburg
  - Boehringer Ingelheim Investigational Site 14, Magdeburg
  - Boehringer Ingelheim Investigational Site 15, Magdeburg
  - Boehringer Ingelheim Investigational Site 16, Magdeburg
  - Boehringer Ingelheim Investigational Site 17, Magdeburg
  - Boehringer Ingelheim Investigational Site 1, Magdeburg
  - Boehringer Ingelheim Investigational Site 2, Magdeburg
  - Boehringer Ingelheim Investigational Site 3, Magdeburg
  - Boehringer Ingelheim Investigational Site 4, Magdeburg
  - Boehringer Ingelheim Investigational Site 5, Magdeburg
  - Boehringer Ingelheim Investigational Site 6, Magdeburg
  - Boehringer Ingelheim Investigational Site 7, Magdeburg
  - Boehringer Ingelheim Investigational Site 8, Magdeburg
  - Boehringer Ingelheim Investigational Site 9, Magdeburg
  - Boehringer Ingelheim Investigational Site, Mainburg
  - Boehringer Ingelheim Investigational Site, Maintal
  - Boehringer Ingelheim Investigational Site 1, Mainz
  - Boehringer Ingelheim Investigational Site 2, Mainz
  - Boehringer Ingelheim Investigational Site, Malchow
  - Boehringer Ingelheim Investigational Site 1, Malente
  - Boehringer Ingelheim Investigational Site 2, Malente
  - Boehringer Ingelheim Investigational Site, Mammendorf
  - Boehringer Ingelheim Investigational Site, Mandelbachtal
  - Boehringer Ingelheim Investigational Site 10, Mannheim
  - Boehringer Ingelheim Investigational Site 11, Mannheim
  - Boehringer Ingelheim Investigational Site 12, Mannheim
  - Boehringer Ingelheim Investigational Site 13, Mannheim
  - Boehringer Ingelheim Investigational Site 14, Mannheim
  - Boehringer Ingelheim Investigational Site 15, Mannheim
  - Boehringer Ingelheim Investigational Site 16, Mannheim
  - Boehringer Ingelheim Investigational Site 1, Mannheim
  - Boehringer Ingelheim Investigational Site 2, Mannheim
  - Boehringer Ingelheim Investigational Site 3, Mannheim
  - Boehringer Ingelheim Investigational Site 4, Mannheim
  - Boehringer Ingelheim Investigational Site 5, Mannheim
  - Boehringer Ingelheim Investigational Site 6, Mannheim
  - Boehringer Ingelheim Investigational Site 7, Mannheim
  - Boehringer Ingelheim Investigational Site 8, Mannheim
  - Boehringer Ingelheim Investigational Site 9, Mannheim
  - Boehringer Ingelheim Investigational Site, Marburg
  - Boehringer Ingelheim Investigational Site, Markersdorf
  - Boehringer Ingelheim Investigational Site, Marklohe
  - Boehringer Ingelheim Investigational Site, Marktheidenfeld
  - Boehringer Ingelheim Investigational Site, Marktleugast
  - Boehringer Ingelheim Investigational Site, Marktoberdorf
  - Boehringer Ingelheim Investigational Site, Marktrodach
  - Boehringer Ingelheim Investigational Site 1, Marl
  - Boehringer Ingelheim Investigational Site 2, Marl
  - Boehringer Ingelheim Investigational Site 3, Marl
  - Boehringer Ingelheim Investigational Site, Marsberg
  - Boehringer Ingelheim Investigational Site, Maulbronn
  - Boehringer Ingelheim Investigational Site, Maulburg
  - Boehringer Ingelheim Investigational Site, Mayen
  - Boehringer Ingelheim Investigational Site 1, Meckenheim
  - Boehringer Ingelheim Investigational Site 2, Meckenheim
  - Boehringer Ingelheim Investigational Site 3, Meckenheim
  - Boehringer Ingelheim Investigational Site, Meerbusch
  - Boehringer Ingelheim Investigational Site, Meinerzhagen
  - Boehringer Ingelheim Investigational Site 1, Meinhard
  - Boehringer Ingelheim Investigational Site 2, Meinhard
  - Boehringer Ingelheim Investigational Site, Meisenheim
  - Boehringer Ingelheim Investigational Site, Meißen
  - Boehringer Ingelheim Investigational Site, Melle
  - Boehringer Ingelheim Investigational Site 1, Mellrichstadt
  - Boehringer Ingelheim Investigational Site 2, Mellrichstadt
  - Boehringer Ingelheim Investigational Site 3, Mellrichstadt
  - Boehringer Ingelheim Investigational Site, Melsungen
  - Boehringer Ingelheim Investigational Site, Memmelsdorf
  - Boehringer Ingelheim Investigational Site 1, Memmingen
  - Boehringer Ingelheim Investigational Site 2, Memmingen
  - Boehringer Ingelheim Investigational Site 1, Menden
  - Boehringer Ingelheim Investigational Site 2, Menden
  - Boehringer Ingelheim Investigational Site, Mendig
  - Boehringer Ingelheim Investigational Site, Menteroda
  - Boehringer Ingelheim Investigational Site, Merchweiler
  - Boehringer Ingelheim Investigational Site, Mering
  - Boehringer Ingelheim Investigational Site, Merkendorf
  - Boehringer Ingelheim Investigational Site 1, Merseburg
  - Boehringer Ingelheim Investigational Site 2, Merseburg
  - Boehringer Ingelheim Investigational Site, Merzig
  - Boehringer Ingelheim Investigational Site, Messkirch
  - Boehringer Ingelheim Investigational Site, Mettingen
  - Boehringer Ingelheim Investigational Site, Mettlach
  - Boehringer Ingelheim Investigational Site, Mettmann
  - Boehringer Ingelheim Investigational Site, Meuselwitz
  - Boehringer Ingelheim Investigational Site, Michelstadt
  - Boehringer Ingelheim Investigational Site, Mildstedt
  - Boehringer Ingelheim Investigational Site, Mindelstetten
  - Boehringer Ingelheim Investigational Site 1, Minden
  - Boehringer Ingelheim Investigational Site 2, Minden
  - Boehringer Ingelheim Investigational Site, Mittenaar
  - Boehringer Ingelheim Investigational Site 1, Mittweida
  - Boehringer Ingelheim Investigational Site 2, Mittweida
  - Boehringer Ingelheim Investigational Site 3, Mittweida
  - Boehringer Ingelheim Investigational Site 1, Moers
  - Boehringer Ingelheim Investigational Site 2, Moers
  - Boehringer Ingelheim Investigational Site 1, Monheim
  - Boehringer Ingelheim Investigational Site 2, Monheim
  - Boehringer Ingelheim Investigational Site, Moormerland
  - Boehringer Ingelheim Investigational Site 10, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 1, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 2, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 3, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 4, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 5, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 6, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 7, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 8, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 9, Mönchengladbach
  - Boehringer Ingelheim Investigational Site, Mönkeberg
  - Boehringer Ingelheim Investigational Site, Mörlenbach
  - Boehringer Ingelheim Investigational Site, Mudersbach
  - Boehringer Ingelheim Investigational Site, Munderkingen
  - Boehringer Ingelheim Investigational Site, Murg
  - Boehringer Ingelheim Investigational Site 1, Mügeln
  - Boehringer Ingelheim Investigational Site 2, Mügeln
  - Boehringer Ingelheim Investigational Site, Mügeln
  - Boehringer Ingelheim Investigational Site 1, Mühlhausen
  - Boehringer Ingelheim Investigational Site 2, Mühlhausen
  - Boehringer Ingelheim Investigational Site 3, Mühlhausen
  - Boehringer Ingelheim Investigational Site 4, Mühlhausen
  - Boehringer Ingelheim Investigational Site 5, Mühlhausen
  - Boehringer Ingelheim Investigational Site 6, Mühlhausen
  - Boehringer Ingelheim Investigational Site 7, Mühlhausen
  - Boehringer Ingelheim Investigational Site 1, Mülheim
  - Boehringer Ingelheim Investigational Site 2, Mülheim
  - Boehringer Ingelheim Investigational Site 3, Mülheim
  - Boehringer Ingelheim Investigational Site 4, Mülheim
  - Boehringer Ingelheim Investigational Site, Münchberg
  - Boehringer Ingelheim Investigational Site, Müncheberg
  - Boehringer Ingelheim Investigational Site 10, München
  - Boehringer Ingelheim Investigational Site 11, München
  - Boehringer Ingelheim Investigational Site 12, München
  - Boehringer Ingelheim Investigational Site 13, München
  - Boehringer Ingelheim Investigational Site 14, München
  - Boehringer Ingelheim Investigational Site 15, München
  - Boehringer Ingelheim Investigational Site 16, München
  - Boehringer Ingelheim Investigational Site 17, München
  - Boehringer Ingelheim Investigational Site 18, München
  - Boehringer Ingelheim Investigational Site 19, München
  - Boehringer Ingelheim Investigational Site 1, München
  - Boehringer Ingelheim Investigational Site 20, München
  - Boehringer Ingelheim Investigational Site 21, München
  - Boehringer Ingelheim Investigational Site 22, München
  - Boehringer Ingelheim Investigational Site 23, München
  - Boehringer Ingelheim Investigational Site 2, München
  - Boehringer Ingelheim Investigational Site 3, München
  - Boehringer Ingelheim Investigational Site 4, München
  - Boehringer Ingelheim Investigational Site 5, München
  - Boehringer Ingelheim Investigational Site 6, München
  - Boehringer Ingelheim Investigational Site 7, München
  - Boehringer Ingelheim Investigational Site 8, München
  - Boehringer Ingelheim Investigational Site 9, München
  - Boehringer Ingelheim Investigational Site, Münchsteinach
  - Boehringer Ingelheim Investigational Site 1, Münster
  - Boehringer Ingelheim Investigational Site 2, Münster
  - Boehringer Ingelheim Investigational Site 3, Münster
  - Boehringer Ingelheim Investigational Site 4, Münster
  - Boehringer Ingelheim Investigational Site 1, Münzenberg
  - Boehringer Ingelheim Investigational Site 2, Münzenberg
  - Boehringer Ingelheim Investigational Site, Nahe
  - Boehringer Ingelheim Investigational Site, Namborn
  - Boehringer Ingelheim Investigational Site, Nandlstadt
  - Boehringer Ingelheim Investigational Site, Nassau
  - Boehringer Ingelheim Investigational Site, Nastätten
  - Boehringer Ingelheim Investigational Site, Nauen
  - Boehringer Ingelheim Investigational Site, Naundorf
  - Boehringer Ingelheim Investigational Site, Neckartailfingen
  - Boehringer Ingelheim Investigational Site, Nellingen
  - Boehringer Ingelheim Investigational Site 1, Netphen
  - Boehringer Ingelheim Investigational Site 2, Netphen
  - Boehringer Ingelheim Investigational Site, Nettersheim
  - Boehringer Ingelheim Investigational Site 1, Nettetal
  - Boehringer Ingelheim Investigational Site 2, Nettetal
  - Boehringer Ingelheim Investigational Site, Neu Kaliß
  - Boehringer Ingelheim Investigational Site, Neu-Isenburg
  - Boehringer Ingelheim Investigational Site, Neu-Ulm
  - Boehringer Ingelheim Investigational Site 1, Neubrandenburg
  - Boehringer Ingelheim Investigational Site 2, Neubrandenburg
  - Boehringer Ingelheim Investigational Site, Neuenkirchen
  - Boehringer Ingelheim Investigational Site, Neuenrade
  - Boehringer Ingelheim Investigational Site, Neugersdorf
  - Boehringer Ingelheim Investigational Site, Neuhaus
  - Boehringer Ingelheim Investigational Site, Neuhof
  - Boehringer Ingelheim Investigational Site, Neuhofen
  - Boehringer Ingelheim Investigational Site 1, Neukirchen
  - Boehringer Ingelheim Investigational Site 2, Neukirchen
  - Boehringer Ingelheim Investigational Site, Neulußheim
  - Boehringer Ingelheim Investigational Site 1, Neumünster
  - Boehringer Ingelheim Investigational Site 2, Neumünster
  - Boehringer Ingelheim Investigational Site 3, Neumünster
  - Boehringer Ingelheim Investigational Site 4, Neumünster
  - Boehringer Ingelheim Investigational Site 1, Neunkirchen
  - Boehringer Ingelheim Investigational Site 2, Neunkirchen
  - Boehringer Ingelheim Investigational Site 1, Neuruppin
  - Boehringer Ingelheim Investigational Site 2, Neuruppin
  - Boehringer Ingelheim Investigational Site 1, Neuss
  - Boehringer Ingelheim Investigational Site 2, Neuss
  - Boehringer Ingelheim Investigational Site 3, Neuss
  - Boehringer Ingelheim Investigational Site 4, Neuss
  - Boehringer Ingelheim Investigational Site 5, Neuss
  - Boehringer Ingelheim Investigational Site 6, Neuss
  - Boehringer Ingelheim Investigational Site 1, Neustadt
  - Boehringer Ingelheim Investigational Site 2, Neustadt
  - Boehringer Ingelheim Investigational Site 3, Neustadt
  - Boehringer Ingelheim Investigational Site 4, Neustadt
  - Boehringer Ingelheim Investigational Site 5, Neustadt
  - Boehringer Ingelheim Investigational Site 1, Neuwied
  - Boehringer Ingelheim Investigational Site 2, Neuwied
  - Boehringer Ingelheim Investigational Site 3, Neuwied
  - Boehringer Ingelheim Investigational Site 1, Nidderau
  - Boehringer Ingelheim Investigational Site 2, Nidderau
  - Boehringer Ingelheim Investigational Site 3, Nidderau
  - Boehringer Ingelheim Investigational Site 4, Nidderau
  - Boehringer Ingelheim Investigational Site, Niederaula
  - Boehringer Ingelheim Investigational Site, Niederfischbach
  - Boehringer Ingelheim Investigational Site, Niederkassel
  - Boehringer Ingelheim Investigational Site, Niederlehme
  - Boehringer Ingelheim Investigational Site, Niedernhausen
  - Boehringer Ingelheim Investigational Site, Niedernwöhren
  - Boehringer Ingelheim Investigational Site, Niederpöllnitz
  - Boehringer Ingelheim Investigational Site, Niederstetten
  - Boehringer Ingelheim Investigational Site, Niederwiesa
  - Boehringer Ingelheim Investigational Site, Niederzissen
  - Boehringer Ingelheim Investigational Site, Niemegk
  - Boehringer Ingelheim Investigational Site 1, Nienburg
  - Boehringer Ingelheim Investigational Site 2, Nienburg
  - Boehringer Ingelheim Investigational Site, Nienstädt
  - Boehringer Ingelheim Investigational Site, Niesky
  - Boehringer Ingelheim Investigational Site, Nittendorf
  - Boehringer Ingelheim Investigational Site, Nordenham
  - Boehringer Ingelheim Investigational Site, Nordhausen
  - Boehringer Ingelheim Investigational Site, Nordheim
  - Boehringer Ingelheim Investigational Site, Nordholz
  - Boehringer Ingelheim Investigational Site, Nordkirchen
  - Boehringer Ingelheim Investigational Site, Nordstemmen
  - Boehringer Ingelheim Investigational Site 1, Nordwalde
  - Boehringer Ingelheim Investigational Site 2, Nordwalde
  - Boehringer Ingelheim Investigational Site, Nossen
  - Boehringer Ingelheim Investigational Site, Notzingen
  - Boehringer Ingelheim Investigational Site, Nördlingen
  - Boehringer Ingelheim Investigational Site 1, Nuremberg
  - Boehringer Ingelheim Investigational Site 2, Nuremberg
  - Boehringer Ingelheim Investigational Site 3, Nuremberg
  - Boehringer Ingelheim Investigational Site 4, Nuremberg
  - Boehringer Ingelheim Investigational Site 5, Nuremberg
  - Boehringer Ingelheim Investigational Site 6, Nuremberg
  - Boehringer Ingelheim Investigational Site 7, Nuremberg
  - Boehringer Ingelheim Investigational Site 8, Nuremberg
  - Boehringer Ingelheim Investigational Site 9, Nuremberg
  - Boehringer Ingelheim Investigational Site, Nusplingen
  - Boehringer Ingelheim Investigational Site 1, Nuthetal
  - Boehringer Ingelheim Investigational Site 2, Nuthetal
  - Boehringer Ingelheim Investigational Site, Nünschweiler
  - Boehringer Ingelheim Investigational Site 1, Nürtingen
  - Boehringer Ingelheim Investigational Site 2, Nürtingen
  - Boehringer Ingelheim Investigational Site, Oberasbach
  - Boehringer Ingelheim Investigational Site, Oberaudorf
  - Boehringer Ingelheim Investigational Site, Oberaula
  - Boehringer Ingelheim Investigational Site, Oberdorla
  - Boehringer Ingelheim Investigational Site, Obergurig
  - Boehringer Ingelheim Investigational Site, Oberhaid
  - Boehringer Ingelheim Investigational Site 1, Oberhausen
  - Boehringer Ingelheim Investigational Site 2, Oberhausen
  - Boehringer Ingelheim Investigational Site 3, Oberhausen
  - Boehringer Ingelheim Investigational Site 4, Oberhausen
  - Boehringer Ingelheim Investigational Site 5, Oberhausen
  - Boehringer Ingelheim Investigational Site 6, Oberhausen
  - Boehringer Ingelheim Investigational Site 7, Oberhausen
  - Boehringer Ingelheim Investigational Site 8, Oberhausen
  - Boehringer Ingelheim Investigational Site 1, Oberkirch
  - Boehringer Ingelheim Investigational Site 2, Oberkirch
  - Boehringer Ingelheim Investigational Site, Oberlungwitz
  - Boehringer Ingelheim Investigational Site, Obermichelbach
  - Boehringer Ingelheim Investigational Site, Obernkirchen
  - Boehringer Ingelheim Investigational Site, Oberried
  - Boehringer Ingelheim Investigational Site, Oberursel
  - Boehringer Ingelheim Investigational Site, Oberwiesenthal
  - Boehringer Ingelheim Investigational Site, Ochtendung
  - Boehringer Ingelheim Investigational Site, Ockenheim
  - Boehringer Ingelheim Investigational Site, Oederan
  - Boehringer Ingelheim Investigational Site, Oelde
  - Boehringer Ingelheim Investigational Site 1, Oelsnitz
  - Boehringer Ingelheim Investigational Site 2, Oelsnitz
  - Boehringer Ingelheim Investigational Site 3, Oelsnitz
  - Boehringer Ingelheim Investigational Site 1, Oer-Erkenschwick
  - Boehringer Ingelheim Investigational Site 2, Oer-Erkenschwick
  - Boehringer Ingelheim Investigational Site 3, Oer-Erkenschwick
  - Boehringer Ingelheim Investigational Site, Oerel
  - Boehringer Ingelheim Investigational Site 1, Offenbach
  - Boehringer Ingelheim Investigational Site 2, Offenbach
  - Boehringer Ingelheim Investigational Site 3, Offenbach
  - Boehringer Ingelheim Investigational Site 4, Offenbach
  - Boehringer Ingelheim Investigational Site, Offstein
  - Boehringer Ingelheim Investigational Site, Olbernhau
  - Boehringer Ingelheim Investigational Site, Olching
  - Boehringer Ingelheim Investigational Site, Oldenburg
  - Boehringer Ingelheim Investigational Site, Oldendorf
  - Boehringer Ingelheim Investigational Site, Oppenheim
  - Boehringer Ingelheim Investigational Site 1, Oranienburg
  - Boehringer Ingelheim Investigational Site 2, Oranienburg
  - Boehringer Ingelheim Investigational Site, Orenhofen
  - Boehringer Ingelheim Investigational Site 1, Oschatz
  - Boehringer Ingelheim Investigational Site 2, Oschatz
  - Boehringer Ingelheim Investigational Site 3, Oschatz
  - Boehringer Ingelheim Investigational Site, Osloß
  - Boehringer Ingelheim Investigational Site 1, Osnabrück
  - Boehringer Ingelheim Investigational Site 2, Osnabrück
  - Boehringer Ingelheim Investigational Site 3, Osnabrück
  - Boehringer Ingelheim Investigational Site, Ostercappeln
  - Boehringer Ingelheim Investigational Site, Osterhausen
  - Boehringer Ingelheim Investigational Site, Osterhofen
  - Boehringer Ingelheim Investigational Site 1, Osterode
  - Boehringer Ingelheim Investigational Site 2, Osterode
  - Boehringer Ingelheim Investigational Site 3, Osterode
  - Boehringer Ingelheim Investigational Site 4, Osterode
  - Boehringer Ingelheim Investigational Site 5, Osterode
  - Boehringer Ingelheim Investigational Site 6, Osterode
  - Boehringer Ingelheim Investigational Site 7, Osterode
  - Boehringer Ingelheim Investigational Site 1, Ostseebad Binz
  - Boehringer Ingelheim Investigational Site 2, Ostseebad Binz
  - Boehringer Ingelheim Investigational Site, Ostseebad Kühlungsborn
  - Boehringer Ingelheim Investigational Site, Otterbach
  - Boehringer Ingelheim Investigational Site, Otterndorf
  - Boehringer Ingelheim Investigational Site, Ottersberg
  - Boehringer Ingelheim Investigational Site, Otterstadt
  - Boehringer Ingelheim Investigational Site, Otterwisch
  - Boehringer Ingelheim Investigational Site, Ottweiler
  - Boehringer Ingelheim Investigational Site, Oy-Mittelberg
  - Boehringer Ingelheim Investigational Site, Öhringen
  - Boehringer Ingelheim Investigational Site 1, Paderborn
  - Boehringer Ingelheim Investigational Site 2, Paderborn
  - Boehringer Ingelheim Investigational Site 1, Papenburg
  - Boehringer Ingelheim Investigational Site 2, Papenburg
  - Boehringer Ingelheim Investigational Site 1, Parchim
  - Boehringer Ingelheim Investigational Site 2, Parchim
  - Boehringer Ingelheim Investigational Site, Passau
  - Boehringer Ingelheim Investigational Site 1, Peine
  - Boehringer Ingelheim Investigational Site 2, Peine
  - Boehringer Ingelheim Investigational Site 3, Peine
  - Boehringer Ingelheim Investigational Site, Peiting
  - Boehringer Ingelheim Investigational Site 1, Petershagen
  - Boehringer Ingelheim Investigational Site 2, Petershagen
  - Boehringer Ingelheim Investigational Site 1, Pfaffenhofen
  - Boehringer Ingelheim Investigational Site 2, Pfaffenhofen
  - Boehringer Ingelheim Investigational Site 1, Pforzheim
  - Boehringer Ingelheim Investigational Site 2, Pforzheim
  - Boehringer Ingelheim Investigational Site 3, Pforzheim
  - Boehringer Ingelheim Investigational Site 4, Pforzheim
  - Boehringer Ingelheim Investigational Site, Pfullingen
  - Boehringer Ingelheim Investigational Site 1, Philippsburg
  - Boehringer Ingelheim Investigational Site 2, Philippsburg
  - Boehringer Ingelheim Investigational Site 3, Philippsburg
  - Boehringer Ingelheim Investigational Site 1, Pirmasens
  - Boehringer Ingelheim Investigational Site 2, Pirmasens
  - Boehringer Ingelheim Investigational Site 1, Pirna
  - Boehringer Ingelheim Investigational Site 2, Pirna
  - Boehringer Ingelheim Investigational Site, Plaidt
  - Boehringer Ingelheim Investigational Site, Plate
  - Boehringer Ingelheim Investigational Site 1, Plauen
  - Boehringer Ingelheim Investigational Site 2, Plauen
  - Boehringer Ingelheim Investigational Site 3, Plauen
  - Boehringer Ingelheim Investigational Site 4, Plauen
  - Boehringer Ingelheim Investigational Site 5, Plauen
  - Boehringer Ingelheim Investigational Site 6, Plauen
  - Boehringer Ingelheim Investigational Site 7, Plauen
  - Boehringer Ingelheim Investigational Site, Plettenberg
  - Boehringer Ingelheim Investigational Site, Pluwig
  - Boehringer Ingelheim Investigational Site 1, Potsdam
  - Boehringer Ingelheim Investigational Site 2, Potsdam
  - Boehringer Ingelheim Investigational Site 3, Potsdam
  - Boehringer Ingelheim Investigational Site 4, Potsdam
  - Boehringer Ingelheim Investigational Site 5, Potsdam
  - Boehringer Ingelheim Investigational Site, Pößneck
  - Boehringer Ingelheim Investigational Site, Preetz
  - Boehringer Ingelheim Investigational Site 1, Premnitz
  - Boehringer Ingelheim Investigational Site 2, Premnitz
  - Boehringer Ingelheim Investigational Site, Prenzlau
  - Boehringer Ingelheim Investigational Site 1, Pulheim
  - Boehringer Ingelheim Investigational Site 2, Pulheim
  - Boehringer Ingelheim Investigational Site, Putbus
  - Boehringer Ingelheim Investigational Site, Püttlingen
  - Boehringer Ingelheim Investigational Site, Quedlinburg
  - Boehringer Ingelheim Investigational Site, Queidersbach
  - Boehringer Ingelheim Investigational Site, Quierschied
  - Boehringer Ingelheim Investigational Site, Rabenau
  - Boehringer Ingelheim Investigational Site 1, Radebeul
  - Boehringer Ingelheim Investigational Site 2, Radebeul
  - Boehringer Ingelheim Investigational Site, Radevormwald
  - Boehringer Ingelheim Investigational Site, Ralingen
  - Boehringer Ingelheim Investigational Site, Randersacker
  - Boehringer Ingelheim Investigational Site, Ranis
  - Boehringer Ingelheim Investigational Site, Ransbach-Baumbach
  - Boehringer Ingelheim Investigational Site 1, Rastatt
  - Boehringer Ingelheim Investigational Site 2, Rastatt
  - Boehringer Ingelheim Investigational Site 1, Rastede
  - Boehringer Ingelheim Investigational Site 2, Rastede
  - Boehringer Ingelheim Investigational Site 3, Rastede
  - Boehringer Ingelheim Investigational Site, Ratekau
  - Boehringer Ingelheim Investigational Site, Ratingen
  - Boehringer Ingelheim Investigational Site, Raubach
  - Boehringer Ingelheim Investigational Site 1, Ravensburg
  - Boehringer Ingelheim Investigational Site 2, Ravensburg
  - Boehringer Ingelheim Investigational Site 3, Ravensburg
  - Boehringer Ingelheim Investigational Site 1, Recklinghausen
  - Boehringer Ingelheim Investigational Site 2, Recklinghausen
  - Boehringer Ingelheim Investigational Site, Rees
  - Boehringer Ingelheim Investigational Site, Regen
  - Boehringer Ingelheim Investigational Site 1, Regensburg
  - Boehringer Ingelheim Investigational Site 2, Regensburg
  - Boehringer Ingelheim Investigational Site 3, Regensburg
  - Boehringer Ingelheim Investigational Site 4, Regensburg
  - Boehringer Ingelheim Investigational Site 5, Regensburg
  - Boehringer Ingelheim Investigational Site, Regis-Breitingen
  - Boehringer Ingelheim Investigational Site, Reichelsheim
  - Boehringer Ingelheim Investigational Site, Reichenbach
  - Boehringer Ingelheim Investigational Site, Reichertshofen
  - Boehringer Ingelheim Investigational Site, Reinfeld
  - Boehringer Ingelheim Investigational Site, Reinheim
  - Boehringer Ingelheim Investigational Site, Rellingen
  - Boehringer Ingelheim Investigational Site 1, Remscheid
  - Boehringer Ingelheim Investigational Site 2, Remscheid
  - Boehringer Ingelheim Investigational Site 3, Remscheid
  - Boehringer Ingelheim Investigational Site 4, Remscheid
  - Boehringer Ingelheim Investigational Site 5, Remscheid
  - Boehringer Ingelheim Investigational Site, Remseck
  - Boehringer Ingelheim Investigational Site, Rendsburg
  - Boehringer Ingelheim Investigational Site, Rethem
  - Boehringer Ingelheim Investigational Site, Rhauderfehn
  - Boehringer Ingelheim Investigational Site 1, Rhaunen
  - Boehringer Ingelheim Investigational Site 2, Rhaunen
  - Boehringer Ingelheim Investigational Site, Rheinbach
  - Boehringer Ingelheim Investigational Site 1, Rheinberg
  - Boehringer Ingelheim Investigational Site 2, Rheinberg
  - Boehringer Ingelheim Investigational Site, Rheine
  - Boehringer Ingelheim Investigational Site, Rheinmünster
  - Boehringer Ingelheim Investigational Site, Ribnitz-Damgarten
  - Boehringer Ingelheim Investigational Site, Ried
  - Boehringer Ingelheim Investigational Site, Rieden
  - Boehringer Ingelheim Investigational Site, Riedlingen
  - Boehringer Ingelheim Investigational Site, Riesa
  - Boehringer Ingelheim Investigational Site 1, Rietberg
  - Boehringer Ingelheim Investigational Site 2, Rietberg
  - Boehringer Ingelheim Investigational Site 1, Rinteln
  - Boehringer Ingelheim Investigational Site 2, Rinteln
  - Boehringer Ingelheim Investigational Site, Rochlitz
  - Boehringer Ingelheim Investigational Site, Rodeberg
  - Boehringer Ingelheim Investigational Site 1, Rodenbach
  - Boehringer Ingelheim Investigational Site 2, Rodenbach
  - Boehringer Ingelheim Investigational Site 1, Rodewisch
  - Boehringer Ingelheim Investigational Site 2, Rodewisch
  - Boehringer Ingelheim Investigational Site, Roetgen
  - Boehringer Ingelheim Investigational Site, Rommerskirchen
  - Boehringer Ingelheim Investigational Site, Ronneburg
  - Boehringer Ingelheim Investigational Site, Ronnenberg
  - Boehringer Ingelheim Investigational Site, Rosenfeld
  - Boehringer Ingelheim Investigational Site, Rosengarten
  - Boehringer Ingelheim Investigational Site, Rosenheim
  - Boehringer Ingelheim Investigational Site, Rositz
  - Boehringer Ingelheim Investigational Site 1, Rostock
  - Boehringer Ingelheim Investigational Site 2, Rostock
  - Boehringer Ingelheim Investigational Site 3, Rostock
  - Boehringer Ingelheim Investigational Site 4, Rostock
  - Boehringer Ingelheim Investigational Site 5, Rostock
  - Boehringer Ingelheim Investigational Site 6, Rostock
  - Boehringer Ingelheim Investigational Site 7, Rostock
  - Boehringer Ingelheim Investigational Site 8, Rostock
  - Boehringer Ingelheim Investigational Site, Rotenburg (Wümme)
  - Boehringer Ingelheim Investigational Site, Rott
  - Boehringer Ingelheim Investigational Site, Rottenburg
  - Boehringer Ingelheim Investigational Site, Roßlau
  - Boehringer Ingelheim Investigational Site, Roßwein
  - Boehringer Ingelheim Investigational Site, Rödermark
  - Boehringer Ingelheim Investigational Site, Rödinghausen
  - Boehringer Ingelheim Investigational Site, Rötha
  - Boehringer Ingelheim Investigational Site, Rudersberg
  - Boehringer Ingelheim Investigational Site, Rugendorf
  - Boehringer Ingelheim Investigational Site, Rüdersdorf
  - Boehringer Ingelheim Investigational Site, Rüsselsheim am Main
  - Boehringer Ingelheim Investigational Site 1, Saarbrücken
  - Boehringer Ingelheim Investigational Site 2, Saarbrücken
  - Boehringer Ingelheim Investigational Site 3, Saarbrücken
  - Boehringer Ingelheim Investigational Site 4, Saarbrücken
  - Boehringer Ingelheim Investigational Site, Saarburg
  - Boehringer Ingelheim Investigational Site 1, Saarlouis
  - Boehringer Ingelheim Investigational Site 2, Saarlouis
  - Boehringer Ingelheim Investigational Site 1, Saint Wendel
  - Boehringer Ingelheim Investigational Site 2, Saint Wendel
  - Boehringer Ingelheim Investigational Site 1, Salzgitter
  - Boehringer Ingelheim Investigational Site 2, Salzgitter
  - Boehringer Ingelheim Investigational Site 3, Salzgitter
  - Boehringer Ingelheim Investigational Site 4, Salzgitter
  - Boehringer Ingelheim Investigational Site, Salzwedel
  - Boehringer Ingelheim Investigational Site, Sankt Englmar
  - Boehringer Ingelheim Investigational Site, Sankt Märgen
  - Boehringer Ingelheim Investigational Site, Sarstedt
  - Boehringer Ingelheim Investigational Site, Sassenberg
  - Boehringer Ingelheim Investigational Site, Schellerten
  - Boehringer Ingelheim Investigational Site, Schernberg
  - Boehringer Ingelheim Investigational Site, Schiffweiler
  - Boehringer Ingelheim Investigational Site, Schildau
  - Boehringer Ingelheim Investigational Site, Schleiden
  - Boehringer Ingelheim Investigational Site, Schleiz
  - Boehringer Ingelheim Investigational Site 1, Schleusingen
  - Boehringer Ingelheim Investigational Site 2, Schleusingen
  - Boehringer Ingelheim Investigational Site, Schlotheim
  - Boehringer Ingelheim Investigational Site, Schloß Holte-Stukenbrok
  - Boehringer Ingelheim Investigational Site, Schmalkalden
  - Boehringer Ingelheim Investigational Site, Schnaittach
  - Boehringer Ingelheim Investigational Site, Schorndorf
  - Boehringer Ingelheim Investigational Site, Schöllkrippen
  - Boehringer Ingelheim Investigational Site, Schönberg
  - Boehringer Ingelheim Investigational Site 1, Schönebeck
  - Boehringer Ingelheim Investigational Site 2, Schönebeck
  - Boehringer Ingelheim Investigational Site 3, Schönebeck
  - Boehringer Ingelheim Investigational Site, Schöneck
  - Boehringer Ingelheim Investigational Site 1, Schönenberg-Kübelberg
  - Boehringer Ingelheim Investigational Site 2, Schönenberg-Kübelberg
  - Boehringer Ingelheim Investigational Site, Schönfeld
  - Boehringer Ingelheim Investigational Site, Schönwald
  - Boehringer Ingelheim Investigational Site, Schöppingen
  - Boehringer Ingelheim Investigational Site 1, Schramberg
  - Boehringer Ingelheim Investigational Site 2, Schramberg
  - Boehringer Ingelheim Investigational Site, Schulzendorf
  - Boehringer Ingelheim Investigational Site 1, Schwalbach
  - Boehringer Ingelheim Investigational Site 2, Schwalbach
  - Boehringer Ingelheim Investigational Site 3, Schwalbach
  - Boehringer Ingelheim Investigational Site 1, Schwalmstadt
  - Boehringer Ingelheim Investigational Site 2, Schwalmstadt
  - Boehringer Ingelheim Investigational Site 1, Schwandorf in Bayern
  - Boehringer Ingelheim Investigational Site 2, Schwandorf in Bayern
  - Boehringer Ingelheim Investigational Site, Schwanewede
  - Boehringer Ingelheim Investigational Site, Schwarzach
  - Boehringer Ingelheim Investigational Site, Schwarzenbach A Wald
  - Boehringer Ingelheim Investigational Site 1, Schwarzenbek
  - Boehringer Ingelheim Investigational Site 2, Schwarzenbek
  - Boehringer Ingelheim Investigational Site 1, Schwarzenberg
  - Boehringer Ingelheim Investigational Site 2, Schwarzenberg
  - Boehringer Ingelheim Investigational Site, Schwarzenbruck
  - Boehringer Ingelheim Investigational Site, Schwäbisch Gmünd
  - Boehringer Ingelheim Investigational Site, Schwäbisch Hall
  - Boehringer Ingelheim Investigational Site, Schwedt
  - Boehringer Ingelheim Investigational Site 1, Schweinfurt
  - Boehringer Ingelheim Investigational Site 2, Schweinfurt
  - Boehringer Ingelheim Investigational Site 3, Schweinfurt
  - Boehringer Ingelheim Investigational Site, Schweitenkirchen
  - Boehringer Ingelheim Investigational Site, Schwelm
  - Boehringer Ingelheim Investigational Site 1, Schwerin
  - Boehringer Ingelheim Investigational Site 2, Schwerin
  - Boehringer Ingelheim Investigational Site 1, Schwerte
  - Boehringer Ingelheim Investigational Site 2, Schwerte
  - Boehringer Ingelheim Investigational Site 3, Schwerte
  - Boehringer Ingelheim Investigational Site 4, Schwerte
  - Boehringer Ingelheim Investigational Site 1, Schwetzingen
  - Boehringer Ingelheim Investigational Site 2, Schwetzingen
  - Boehringer Ingelheim Investigational Site, Schwieberdingen
  - Boehringer Ingelheim Investigational Site, Sebnitz
  - Boehringer Ingelheim Investigational Site, Seebach
  - Boehringer Ingelheim Investigational Site, Seeg
  - Boehringer Ingelheim Investigational Site, Seelbach
  - Boehringer Ingelheim Investigational Site, Seelze
  - Boehringer Ingelheim Investigational Site, Selb
  - Boehringer Ingelheim Investigational Site, Sendenhorst
  - Boehringer Ingelheim Investigational Site, Senftenberg
  - Boehringer Ingelheim Investigational Site, Sickte
  - Boehringer Ingelheim Investigational Site 1, Siegen
  - Boehringer Ingelheim Investigational Site 2, Siegen
  - Boehringer Ingelheim Investigational Site 3, Siegen
  - Boehringer Ingelheim Investigational Site, Siersleben
  - Boehringer Ingelheim Investigational Site, Silberhausen
  - Boehringer Ingelheim Investigational Site 1, Simmerath
  - Boehringer Ingelheim Investigational Site 2, Simmerath
  - Boehringer Ingelheim Investigational Site 1, Sindelfingen
  - Boehringer Ingelheim Investigational Site 2, Sindelfingen
  - Boehringer Ingelheim Investigational Site 3, Sindelfingen
  - Boehringer Ingelheim Investigational Site 4, Sindelfingen
  - Boehringer Ingelheim Investigational Site 1, Singen
  - Boehringer Ingelheim Investigational Site 2, Singen
  - Boehringer Ingelheim Investigational Site, Singhofen
  - Boehringer Ingelheim Investigational Site 1, Solingen
  - Boehringer Ingelheim Investigational Site 2, Solingen
  - Boehringer Ingelheim Investigational Site 3, Solingen
  - Boehringer Ingelheim Investigational Site 4, Solingen
  - Boehringer Ingelheim Investigational Site 5, Solingen
  - Boehringer Ingelheim Investigational Site 6, Solingen
  - Boehringer Ingelheim Investigational Site 7, Solingen
  - Boehringer Ingelheim Investigational Site, Soltau
  - Boehringer Ingelheim Investigational Site, Sommerach
  - Boehringer Ingelheim Investigational Site 1, Sonneberg
  - Boehringer Ingelheim Investigational Site 2, Sonneberg
  - Boehringer Ingelheim Investigational Site, Sonsbeck
  - Boehringer Ingelheim Investigational Site, Sögel
  - Boehringer Ingelheim Investigational Site, Söhlde
  - Boehringer Ingelheim Investigational Site, Spangenberg
  - Boehringer Ingelheim Investigational Site, Speicher
  - Boehringer Ingelheim Investigational Site, Speichersdorf
  - Boehringer Ingelheim Investigational Site, Spelle
  - Boehringer Ingelheim Investigational Site 1, Speyer
  - Boehringer Ingelheim Investigational Site 2, Speyer
  - Boehringer Ingelheim Investigational Site, Spremberg
  - Boehringer Ingelheim Investigational Site, Springe
  - Boehringer Ingelheim Investigational Site 1, Sprockhövel
  - Boehringer Ingelheim Investigational Site 2, Sprockhövel
  - Boehringer Ingelheim Investigational Site, St. Peter
  - Boehringer Ingelheim Investigational Site 1, Stadland
  - Boehringer Ingelheim Investigational Site 2, Stadland
  - Boehringer Ingelheim Investigational Site, Stadtallendorf
  - Boehringer Ingelheim Investigational Site 1, Stadthagen
  - Boehringer Ingelheim Investigational Site 2, Stadthagen
  - Boehringer Ingelheim Investigational Site 3, Stadthagen
  - Boehringer Ingelheim Investigational Site 4, Stadthagen
  - Boehringer Ingelheim Investigational Site, Stadtlengsfeld
  - Boehringer Ingelheim Investigational Site 1, Stadtlohn
  - Boehringer Ingelheim Investigational Site 2, Stadtlohn
  - Boehringer Ingelheim Investigational Site, Stadtsteinach
  - Boehringer Ingelheim Investigational Site, Stahnsdorf
  - Boehringer Ingelheim Investigational Site, Stamsried
  - Boehringer Ingelheim Investigational Site, Starkenberg
  - Boehringer Ingelheim Investigational Site 1, Staufenberg
  - Boehringer Ingelheim Investigational Site 2, Staufenberg
  - Boehringer Ingelheim Investigational Site 1, Staßfurt
  - Boehringer Ingelheim Investigational Site 2, Staßfurt
  - Boehringer Ingelheim Investigational Site 3, Staßfurt
  - Boehringer Ingelheim Investigational Site 4, Staßfurt
  - Boehringer Ingelheim Investigational Site, Steimel
  - Boehringer Ingelheim Investigational Site, Steinfeld
  - Boehringer Ingelheim Investigational Site, Steinfurt
  - Boehringer Ingelheim Investigational Site, Steinheid
  - Boehringer Ingelheim Investigational Site, Steinmauern
  - Boehringer Ingelheim Investigational Site, Steinwiesen
  - Boehringer Ingelheim Investigational Site 1, Stendal
  - Boehringer Ingelheim Investigational Site 2, Stendal
  - Boehringer Ingelheim Investigational Site 1, Sternberg
  - Boehringer Ingelheim Investigational Site 2, Sternberg
  - Boehringer Ingelheim Investigational Site, Stolberg
  - Boehringer Ingelheim Investigational Site, Stolzenau
  - Boehringer Ingelheim Investigational Site, Storkow
  - Boehringer Ingelheim Investigational Site, Straelen
  - Boehringer Ingelheim Investigational Site, Stralsund
  - Boehringer Ingelheim Investigational Site, Strausberg
  - Boehringer Ingelheim Investigational Site, Straßkirchen
  - Boehringer Ingelheim Investigational Site, Stuhr
  - Boehringer Ingelheim Investigational Site, Stutensee
  - Boehringer Ingelheim Investigational Site 1, Stuttgart
  - Boehringer Ingelheim Investigational Site 2, Stuttgart
  - Boehringer Ingelheim Investigational Site 3, Stuttgart
  - Boehringer Ingelheim Investigational Site 4, Stuttgart
  - Boehringer Ingelheim Investigational Site 5, Stuttgart
  - Boehringer Ingelheim Investigational Site 6, Stuttgart
  - Boehringer Ingelheim Investigational Site 7, Stuttgart
  - Boehringer Ingelheim Investigational Site 8, Stuttgart
  - Boehringer Ingelheim Investigational Site 1, Suhl
  - Boehringer Ingelheim Investigational Site 2, Suhl
  - Boehringer Ingelheim Investigational Site 3, Suhl
  - Boehringer Ingelheim Investigational Site, Sulzbach-Rosenberg
  - Boehringer Ingelheim Investigational Site, Sundern
  - Boehringer Ingelheim Investigational Site, Südbrookmerland
  - Boehringer Ingelheim Investigational Site, Süderbrarup
  - Boehringer Ingelheim Investigational Site, Tanna
  - Boehringer Ingelheim Investigational Site, Teisendorf
  - Boehringer Ingelheim Investigational Site, Teising
  - Boehringer Ingelheim Investigational Site, Teistungen
  - Boehringer Ingelheim Investigational Site 1, Teltow
  - Boehringer Ingelheim Investigational Site 2, Teltow
  - Boehringer Ingelheim Investigational Site 3, Teltow
  - Boehringer Ingelheim Investigational Site, Teutschenthal
  - Boehringer Ingelheim Investigational Site, Thale
  - Boehringer Ingelheim Investigational Site, Thallwitz
  - Boehringer Ingelheim Investigational Site, Thurnau
  - Boehringer Ingelheim Investigational Site 1, Tiefenort
  - Boehringer Ingelheim Investigational Site 2, Tiefenort
  - Boehringer Ingelheim Investigational Site, Tirpersdorf
  - Boehringer Ingelheim Investigational Site, Tirschenreuth
  - Boehringer Ingelheim Investigational Site, Tittling
  - Boehringer Ingelheim Investigational Site, Titz
  - Boehringer Ingelheim Investigational Site, Tönisvorst
  - Boehringer Ingelheim Investigational Site, Trappenkamp
  - Boehringer Ingelheim Investigational Site, Traunreut
  - Boehringer Ingelheim Investigational Site 1, Trebbin
  - Boehringer Ingelheim Investigational Site 2, Trebbin
  - Boehringer Ingelheim Investigational Site, Treis-Karden
  - Boehringer Ingelheim Investigational Site 1, Treuchtlingen
  - Boehringer Ingelheim Investigational Site, Treuchtlingen
  - Boehringer Ingelheim Investigational Site 1, Trier
  - Boehringer Ingelheim Investigational Site 2, Trier
  - Boehringer Ingelheim Investigational Site 1, Triptis
  - Boehringer Ingelheim Investigational Site 2, Triptis
  - Boehringer Ingelheim Investigational Site 3, Triptis
  - Boehringer Ingelheim Investigational Site, Uchte
  - Boehringer Ingelheim Investigational Site, Ueckermünde
  - Boehringer Ingelheim Investigational Site, Uetze
  - Boehringer Ingelheim Investigational Site, Uichteritz
  - Boehringer Ingelheim Investigational Site 1, Ulm
  - Boehringer Ingelheim Investigational Site 2, Ulm
  - Boehringer Ingelheim Investigational Site 1, Undenheim
  - Boehringer Ingelheim Investigational Site 2, Undenheim
  - Boehringer Ingelheim Investigational Site, Unkel
  - Boehringer Ingelheim Investigational Site 1, Unna
  - Boehringer Ingelheim Investigational Site 2, Unna
  - Boehringer Ingelheim Investigational Site 3, Unna
  - Boehringer Ingelheim Investigational Site, Unterlüß
  - Boehringer Ingelheim Investigational Site, Unterschneidheim
  - Boehringer Ingelheim Investigational Site, Untersiemau
  - Boehringer Ingelheim Investigational Site, Unterspreewald
  - Boehringer Ingelheim Investigational Site, Unterwellenborn
  - Boehringer Ingelheim Investigational Site 1, Urbach
  - Boehringer Ingelheim Investigational Site 2, Urbach
  - Boehringer Ingelheim Investigational Site 3, Urbach
  - Boehringer Ingelheim Investigational Site 1, Übach-Palenberg
  - Boehringer Ingelheim Investigational Site 2, Übach-Palenberg
  - Boehringer Ingelheim Investigational Site, Überlingen
  - Boehringer Ingelheim Investigational Site, Ühlingen-Birkendorf
  - Boehringer Ingelheim Investigational Site, Vallendar
  - Boehringer Ingelheim Investigational Site, Vechelde
  - Boehringer Ingelheim Investigational Site, Vechta
  - Boehringer Ingelheim Investigational Site, Veilsdorf
  - Boehringer Ingelheim Investigational Site 1, Velen
  - Boehringer Ingelheim Investigational Site 2, Velen
  - Boehringer Ingelheim Investigational Site, Velten
  - Boehringer Ingelheim Investigational Site 1, Veringenstadt
  - Boehringer Ingelheim Investigational Site 2, Veringenstadt
  - Boehringer Ingelheim Investigational Site, Versmold
  - Boehringer Ingelheim Investigational Site, Vettelschoß
  - Boehringer Ingelheim Investigational Site, Viernau
  - Boehringer Ingelheim Investigational Site 1, Viernheim
  - Boehringer Ingelheim Investigational Site 2, Viernheim
  - Boehringer Ingelheim Investigational Site 3, Viernheim
  - Boehringer Ingelheim Investigational Site 1, Viersen
  - Boehringer Ingelheim Investigational Site 2, Viersen
  - Boehringer Ingelheim Investigational Site 3, Viersen
  - Boehringer Ingelheim Investigational Site, Villingen-Schwenningen
  - Boehringer Ingelheim Investigational Site 1, Vilshofen
  - Boehringer Ingelheim Investigational Site 2, Vilshofen
  - Boehringer Ingelheim Investigational Site 3, Vilshofen
  - Boehringer Ingelheim Investigational Site 1, Visselhövede
  - Boehringer Ingelheim Investigational Site 2, Visselhövede
  - Boehringer Ingelheim Investigational Site, Vitzenburg
  - Boehringer Ingelheim Investigational Site, Vohburg an der Donau
  - Boehringer Ingelheim Investigational Site, Vöhl
  - Boehringer Ingelheim Investigational Site, Vöhrenbach
  - Boehringer Ingelheim Investigational Site 1, Völklingen
  - Boehringer Ingelheim Investigational Site 2, Völklingen
  - Boehringer Ingelheim Investigational Site, Wachtendonk
  - Boehringer Ingelheim Investigational Site, Wadern
  - Boehringer Ingelheim Investigational Site, Wadgassen
  - Boehringer Ingelheim Investigational Site, Wahlstedt
  - Boehringer Ingelheim Investigational Site, Wald-Michelbach
  - Boehringer Ingelheim Investigational Site 1, Waldbreitbach
  - Boehringer Ingelheim Investigational Site 2, Waldbreitbach
  - Boehringer Ingelheim Investigational Site, Waldbrunn
  - Boehringer Ingelheim Investigational Site, Waldkraiburg
  - Boehringer Ingelheim Investigational Site, Waldshut-Tiengen
  - Boehringer Ingelheim Investigational Site, Wallerfing
  - Boehringer Ingelheim Investigational Site, Walzbachtal
  - Boehringer Ingelheim Investigational Site, Wangen
  - Boehringer Ingelheim Investigational Site, Wangerland
  - Boehringer Ingelheim Investigational Site, Wankendorf
  - Boehringer Ingelheim Investigational Site, Wannweil
  - Boehringer Ingelheim Investigational Site, Wardenburg
  - Boehringer Ingelheim Investigational Site 1, Warendorf
  - Boehringer Ingelheim Investigational Site 2, Warendorf
  - Boehringer Ingelheim Investigational Site 1, Warstein
  - Boehringer Ingelheim Investigational Site 2, Warstein
  - Boehringer Ingelheim Investigational Site, Wedel
  - Boehringer Ingelheim Investigational Site, Wedemark
  - Boehringer Ingelheim Investigational Site 1, Weener
  - Boehringer Ingelheim Investigational Site 2, Weener
  - Boehringer Ingelheim Investigational Site, Wehr
  - Boehringer Ingelheim Investigational Site, Weibern
  - Boehringer Ingelheim Investigational Site, Weida
  - Boehringer Ingelheim Investigational Site, Weidenbach
  - Boehringer Ingelheim Investigational Site, Weil am Rhein
  - Boehringer Ingelheim Investigational Site 1, Weimar
  - Boehringer Ingelheim Investigational Site 2, Weimar
  - Boehringer Ingelheim Investigational Site, Weinbergen
  - Boehringer Ingelheim Investigational Site, Weinböhla
  - Boehringer Ingelheim Investigational Site, Weingarten
  - Boehringer Ingelheim Investigational Site, Weinheim
  - Boehringer Ingelheim Investigational Site, Weiskirchen
  - Boehringer Ingelheim Investigational Site, Weissensee
  - Boehringer Ingelheim Investigational Site, Weißenberg
  - Boehringer Ingelheim Investigational Site, Weißenburg
  - Boehringer Ingelheim Investigational Site, Weißenstadt
  - Boehringer Ingelheim Investigational Site, Weißwasser
  - Boehringer Ingelheim Investigational Site, Welschneudorf
  - Boehringer Ingelheim Investigational Site, Welver
  - Boehringer Ingelheim Investigational Site, Welzheim
  - Boehringer Ingelheim Investigational Site, Wemding
  - Boehringer Ingelheim Investigational Site, Wendelstein
  - Boehringer Ingelheim Investigational Site, Wennigsen
  - Boehringer Ingelheim Investigational Site 1, Wermelskirchen
  - Boehringer Ingelheim Investigational Site 2, Wermelskirchen
  - Boehringer Ingelheim Investigational Site, Wermsdorf
  - Boehringer Ingelheim Investigational Site 1, Werne
  - Boehringer Ingelheim Investigational Site 2, Werne
  - Boehringer Ingelheim Investigational Site 1, Wernigerode
  - Boehringer Ingelheim Investigational Site 2, Wernigerode
  - Boehringer Ingelheim Investigational Site, Wertheim am Main
  - Boehringer Ingelheim Investigational Site 1, Wesel
  - Boehringer Ingelheim Investigational Site 2, Wesel
  - Boehringer Ingelheim Investigational Site 3, Wesel
  - Boehringer Ingelheim Investigational Site 1, Wesseling
  - Boehringer Ingelheim Investigational Site 2, Wesseling
  - Boehringer Ingelheim Investigational Site, Westerkappeln
  - Boehringer Ingelheim Investigational Site, Westerstede
  - Boehringer Ingelheim Investigational Site, Wettenberg
  - Boehringer Ingelheim Investigational Site, Wetter
  - Boehringer Ingelheim Investigational Site, Wettstetten
  - Boehringer Ingelheim Investigational Site 1, Wetzlar
  - Boehringer Ingelheim Investigational Site 2, Wetzlar
  - Boehringer Ingelheim Investigational Site 1, Weyhe
  - Boehringer Ingelheim Investigational Site 2, Weyhe
  - Boehringer Ingelheim Investigational Site, Wickede
  - Boehringer Ingelheim Investigational Site, Wiedensahl
  - Boehringer Ingelheim Investigational Site, Wiefelstede
  - Boehringer Ingelheim Investigational Site, Wiehl
  - Boehringer Ingelheim Investigational Site, Wiernsheim
  - Boehringer Ingelheim Investigational Site, Wiesau
  - Boehringer Ingelheim Investigational Site 10, Wiesbaden
  - Boehringer Ingelheim Investigational Site 1, Wiesbaden
  - Boehringer Ingelheim Investigational Site 2, Wiesbaden
  - Boehringer Ingelheim Investigational Site 3, Wiesbaden
  - Boehringer Ingelheim Investigational Site 4, Wiesbaden
  - Boehringer Ingelheim Investigational Site 5, Wiesbaden
  - Boehringer Ingelheim Investigational Site 6, Wiesbaden
  - Boehringer Ingelheim Investigational Site 7, Wiesbaden
  - Boehringer Ingelheim Investigational Site 8, Wiesbaden
  - Boehringer Ingelheim Investigational Site 9, Wiesbaden
  - Boehringer Ingelheim Investigational Site 1, Wiesloch
  - Boehringer Ingelheim Investigational Site 2, Wiesloch
  - Boehringer Ingelheim Investigational Site 3, Wiesloch
  - Boehringer Ingelheim Investigational Site, Wiesthal
  - Boehringer Ingelheim Investigational Site, Wietzen
  - Boehringer Ingelheim Investigational Site, Wiggensbach
  - Boehringer Ingelheim Investigational Site, Wilburgstetten
  - Boehringer Ingelheim Investigational Site, Wilhelmsfeld
  - Boehringer Ingelheim Investigational Site, Wilhelmshaven
  - Boehringer Ingelheim Investigational Site 1, Wilhermsdorf
  - Boehringer Ingelheim Investigational Site 2, Wilhermsdorf
  - Boehringer Ingelheim Investigational Site, Willebadessen
  - Boehringer Ingelheim Investigational Site, Willich
  - Boehringer Ingelheim Investigational Site, Wilthen
  - Boehringer Ingelheim Investigational Site, Winden
  - Boehringer Ingelheim Investigational Site, Winkelhaid
  - Boehringer Ingelheim Investigational Site, Winsen
  - Boehringer Ingelheim Investigational Site, Wipperfürth
  - Boehringer Ingelheim Investigational Site 1, Wismar
  - Boehringer Ingelheim Investigational Site 2, Wismar
  - Boehringer Ingelheim Investigational Site 3, Wismar
  - Boehringer Ingelheim Investigational Site 1, Witten
  - Boehringer Ingelheim Investigational Site 2, Witten
  - Boehringer Ingelheim Investigational Site 3, Witten
  - Boehringer Ingelheim Investigational Site 4, Witten
  - Boehringer Ingelheim Investigational Site 5, Witten
  - Boehringer Ingelheim Investigational Site 1, Wittenberg
  - Boehringer Ingelheim Investigational Site 2, Wittenberg
  - Boehringer Ingelheim Investigational Site, Wittgensdorf
  - Boehringer Ingelheim Investigational Site 1, Wittstock
  - Boehringer Ingelheim Investigational Site 2, Wittstock
  - Boehringer Ingelheim Investigational Site 1, Witzenhausen
  - Boehringer Ingelheim Investigational Site 2, Witzenhausen
  - Boehringer Ingelheim Investigational Site, Wolfen
  - Boehringer Ingelheim Investigational Site, Wolfenbüttel
  - Boehringer Ingelheim Investigational Site 1, Wolfsburg
  - Boehringer Ingelheim Investigational Site 2, Wolfsburg
  - Boehringer Ingelheim Investigational Site 3, Wolfsburg
  - Boehringer Ingelheim Investigational Site 4, Wolfsburg
  - Boehringer Ingelheim Investigational Site 5, Wolfsburg
  - Boehringer Ingelheim Investigational Site 6, Wolfsburg
  - Boehringer Ingelheim Investigational Site 7, Wolfsburg
  - Boehringer Ingelheim Investigational Site 8, Wolfsburg
  - Boehringer Ingelheim Investigational Site, Wolgast
  - Boehringer Ingelheim Investigational Site, Wolmirstedt
  - Boehringer Ingelheim Investigational Site, Wolnzach
  - Boehringer Ingelheim Investigational Site, Worms
  - Boehringer Ingelheim Investigational Site, Wöbbelin
  - Boehringer Ingelheim Investigational Site, Wölfersheim
  - Boehringer Ingelheim Investigational Site, Wöllstein
  - Boehringer Ingelheim Investigational Site 1, Wörrstadt
  - Boehringer Ingelheim Investigational Site 2, Wörrstadt
  - Boehringer Ingelheim Investigational Site 1, Wörth
  - Boehringer Ingelheim Investigational Site 2, Wörth
  - Boehringer Ingelheim Investigational Site, Wriezen
  - Boehringer Ingelheim Investigational Site 1, Wuppertal
  - Boehringer Ingelheim Investigational Site 2, Wuppertal
  - Boehringer Ingelheim Investigational Site 3, Wuppertal
  - Boehringer Ingelheim Investigational Site 4, Wuppertal
  - Boehringer Ingelheim Investigational Site 5, Wuppertal
  - Boehringer Ingelheim Investigational Site, Wustermark
  - Boehringer Ingelheim Investigational Site, Wustrau
  - Boehringer Ingelheim Investigational Site 1, Würselen
  - Boehringer Ingelheim Investigational Site 2, Würselen
  - Boehringer Ingelheim Investigational Site 1, Würzburg
  - Boehringer Ingelheim Investigational Site 2, Würzburg
  - Boehringer Ingelheim Investigational Site 3, Würzburg
  - Boehringer Ingelheim Investigational Site 4, Würzburg
  - Boehringer Ingelheim Investigational Site 1, Xanten
  - Boehringer Ingelheim Investigational Site 2, Xanten
  - Boehringer Ingelheim Investigational Site 1, Zapfendorf
  - Boehringer Ingelheim Investigational Site 2, Zapfendorf
  - Boehringer Ingelheim Investigational Site, Zeesen
  - Boehringer Ingelheim Investigational Site, Zeitz
  - Boehringer Ingelheim Investigational Site 1, Zell
  - Boehringer Ingelheim Investigational Site 2, Zell
  - Boehringer Ingelheim Investigational Site 1, Zerbst
  - Boehringer Ingelheim Investigational Site 2, Zerbst
  - Boehringer Ingelheim Investigational Site, Zernitz
  - Boehringer Ingelheim Investigational Site, Ziltendorf
  - Boehringer Ingelheim Investigational Site, Zingst
  - Boehringer Ingelheim Investigational Site, Zittau
  - Boehringer Ingelheim Investigational Site, Zörbig
  - Boehringer Ingelheim Investigational Site, Zschepplin
  - Boehringer Ingelheim Investigational Site 1, Zschopau
  - Boehringer Ingelheim Investigational Site 2, Zschopau
  - Boehringer Ingelheim Investigational Site, Zulpich
  - Boehringer Ingelheim Investigational Site, Zwenkau
  - Boehringer Ingelheim Investigational Site 1, Zwickau
  - Boehringer Ingelheim Investigational Site 2, Zwickau
  - Boehringer Ingelheim Investigational Site 3, Zwickau
  - Boehringer Ingelheim Investigational Site 4, Zwickau
  - Boehringer Ingelheim Investigational Site 5, Zwickau
  - Boehringer Ingelheim Investigational Site 6, Zwickau
  - Boehringer Ingelheim Investigational Site 7, Zwickau